A Multicenter, Partially-Masked, Randomized, Controlled Study of Medical Therapy vs.
Medical Therapy plus Optic Nerve Sheath Fenestration vs. Medical Therapy plus
Stereotactic Ventriculoperitoneal Cerebrospinal Fluid Shunting in Subjects with Idiopathic
Intracranial Hypertension and Moderate to Severe Visual Loss

Surgical Idiopathic Intracranial Hypertension Treatment Trial ("SIGHT")

IND Sponsor: Michael Wall, MD

Version Number: 4.0

11 April 2019

#### CONFIDENTIAL

This document is a confidential communication of the NORDIC Study Group. The recipient agrees that no information contained herein will be published or disclosed without written approval. This document may be disclosed to appropriate institutional review boards, independent ethics committees, or duly authorized representatives of the U.S. Food & Drug Administration, the Bureau of Pharmaceutical Assessment (Canada), or other regulatory authorities as appropriate; under the condition that confidentiality is requested.

## **KEY ROLES**

| Name, degree | Michael Wall, MD |
|------------------|------------------------------------------|
| Title | Study Director |
| Institution Name | University of Iowa Hospitals and Clinics |
| Name, degree | Matthew Thurtell, MBBS, MSc |
| Title | Study co-Director |
| Institution Name | University of Iowa Hospitals and Clinics |
| Name, degree | Mark Kupersmith, MD |
| Title | Enrollment and Resource Centers Director |
| Institution Name | Mount Sinai |
| Name, degree | Stephanie DuBose, MPH |
| Title | Coordinator Center Director |
| Institution Name | Jaeb Center for Health Research (JCHR) |
| Name, degree | Robert Lindblad, MD |
| Title | Medical Monitor |
| Institution Name | EMMES Corporation |

## **VERSION HISTORY**

The following table lists versions of the protocol:

| VERSION<br>NUMBER | AUTHOR | APPROVER | EFFECTIVE<br>DATE | REVISION DESCRIPTION |
|---|---|---|---|---|
| 1.0 | Michael Wall,<br>Matthew Thurtell,<br>Stephanie<br>DuBose | Stephanie<br>DuBose | 04Jan2018 | Original version |
| 2.0 | Stephanie<br>DuBose | Stephanie<br>DuBose | 20Feb2018 | <ul> <li>Removed terms 'maximal' and 'initial' in reference to medical therapy and clarified that diet is part of medical therapy for all groups</li> <li>Replaced 'study/non-study' eye with 'eligible/non-eligible' eye throughout</li> <li>Modified lumbar puncture inclusion criteria to not require a repeat lumbar puncture if done within 6 weeks (instead of 28 days) and to not require grade II to V papilledema</li> <li>Removed 200-mile inclusion criteria and instead added criteria of good candidate for study based on investigator judgement</li> <li>Added note that if neurologic exam abnormalities are found, the patient should be discussed with the Study Director to determine eligibility</li> <li>Clarification on exclusion criterion for abnormal CT or MRI</li> <li>Removed breastfeeding as exclusion criterion</li> <li>Clarification on how visual field examinations are determined to be reliable and when they will be repeated</li> <li>Removed assessment of furosemide compliance by pill counts since not feasible</li> <li>Removed CBC and Metabolic Panel from study visit procedures at 4 and 8 weeks</li> <li>Clarified that Adjudication Committee will be masked to treatment group and all cases will be reviewed first by the Study Director.</li> <li>Added details on treatment failure criteria and moved surgery specific criteria to appropriate section</li> <li>Clarification on discontinuation of study drug in relation to pregnancy, birth control, and breastfeeding</li> <li>Removed details related to certification of study surgeons, as this will be detailed in the MOP</li> <li>Clarified primary outcome throughout</li> <li>Added clarifications and revisions to statistical chapter</li> <li>Corrected typos</li> </ul> |
| 2.1 | Stephanie<br>DuBose | Stephanie<br>DuBose | 19Mar2018 | <ul> <li>Revised SMRC criteria (text and figure)</li> <li>Updated study design figure to match primary outcome</li> <li>Corrected typos and clarified text throughout</li> <li>Removed extraneous text throughout</li> </ul> |

| VERSION<br>NUMBER | AUTHOR | APPROVER | EFFECTIVE<br>DATE | REVISION DESCRIPTION |
|---|---|---|---|---|
| 2.2 | Stephane<br>DuBose | Stephanie<br>DuBose | 04Apr2018 | <ul> <li>Revised titration and tapering schedule</li> <li>Clarified when to contact Study Director vs co-Director for questions</li> <li>Clarified management of non-eligible eye section to be consistent with rest of protocol</li> <li>Removed specification on timing of repeat perimetry</li> </ul> |
| 3.0 | Stephanie<br>DuBose | Stephanie<br>DuBose | 21May2018 | <ul> <li>Exclusion criterion related to abnormal CSF contents changed to &gt;8 cells, as 0-8 cells in CSF is considered within normal limits</li> <li>Clarified refractive error exclusion</li> <li>Updated AE reporting for known side effects of study drug and surgical AEs</li> <li>Updated details in Stored Specimens section and removed future testing that will not be done; removed duplicate text from data collection chapter</li> <li>Corrected typos</li> <li>Removed unnecessary abbreviations</li> </ul> |
| 3.1 | Stephanie<br>DuBose | Stephanie<br>DuBose | 09Jul2018 | <ul> <li>Amended exclusion criterion related to abnormal CSF contents</li> <li>Corrected typos</li> </ul> |
| 3.2 | Stephanie<br>DuBose | Stephanie<br>DuBose | 23Jul2018 | <ul><li>Updated AE reporting for lab abnormalities</li><li>Corrected typos</li></ul> |
| 4.0 | Nicole Foster,<br>Stephanie<br>DuBose | Stephanie<br>DuBose | 11Apr2019 | <ul> <li>Revised exclusion criteria to allow greater monthly dosage of previous treatment with acetazolamide and methazolamide</li> <li>Revised exclusion criteria regarding conditions requiring steroid use and clarified that during study, steroids only permitted during ONSF surgery.</li> <li>Removed IOP requirement from follow up visits</li> <li>Clarified that size III VF test is optional at screening and not required at 26-week visit</li> <li>Updated amount of blood to be drawn for future research from 50 to 20 ml</li> <li>Revised OCT testing frequency at screening to only be required once instead of twice for all subjects</li> <li>Removed details on tapering schedule for participants in VPS group after shunt, to include in MOP instead</li> <li>Made clarifications to study procedures grid</li> <li>Clarified AE relatedness description to include all study procedures</li> <li>Revised a few analyses details in Statistical Considerations chapter to match Statistical Analysis Plan</li> <li>Corrected typos</li> </ul> |

## TABLE OF CONTENTS

| KEY ROLES | 2 |
|---|---|
| VERSION HISTORY | 3 |
| TABLE OF CONTENTS | 5 |
| LIST OF ABBREVIATIONS | 10 |
| PROTOCOL SUMMARY | 11 |
| CHAPTER 1: INTRODUCTION | 16 |
| 1.1 Background | 16 |
| 1.2 Clinical Experience. | 17 |
| 1.2.1 Visual Loss in IIH | 17 |
| 1.2.2 Optic Nerve Sheath Fenestration for IIH | 17 |
| 1.2.3 CSF Shunting for IIH | 18 |
| 1.2.4 Pilot Data for Management of Moderate to Severe Visual Loss in IIH | 19 |
| 1.2.5 Use of OCT in Monitoring Papilledema in IIH | |
| 1.3 Rationale | 20 |
| 1.3.1 Discussion of Study Design. | 20 |
| 1.3.1.1 Visual Field Monitoring. | 20 |
| 1.3.1.2 OCT Monitoring | 21 |
| 1.3.1.3 Discussion of Subject Characteristics | 22 |
| 1.3.2 Rationale for Medical and Surgical Treatment | 23 |
| 1.3.2.1 Medical Therapy | 23 |
| 1.3.2.2 Optic Nerve Sheath Fenestration | 24 |
| 1.3.2.3 CSF Shunting | 25 |
| 1.4 Study Objectives | 26 |
| 1.4.1 Primary Objective | 26 |
| 1.4.2 Secondary Objectives | 26 |
| 1.4.3 Other Outcomes | 27 |
| 1.5 Potential Risks and Benefits of the Study Interventions | 27 |
| 1.5.1 Known Potential Risks | 27 |
| 1.5.1.1 Visual Loss | 27 |
| 1.5.1.2 Acetazolamide | 27 |
| 1.5.1.3 Furosemide | 28 |
| 1.5.2 Known Potential Benefits | 28 |

| 1.5.3 Risk Assessment | 28 |
|-------------------------------------------------------------|----|
| 1.6 General Considerations | 29 |
| 1.7 Schematic of Study Design | 29 |
| 1.8 Schedule of Study Visits and Procedures | 30 |
| 1.8.1 Randomized Trial | 30 |
| 1.8.2 Treatment Failure Identification Phase | 32 |
| CHAPTER 2: STUDY ENROLLMENT AND SCREENING/BASELINE TESTING | 33 |
| 2.1 Subject Recruitment and Enrollment | |
| 2.1.1 Informed Consent and Authorization Procedures | |
| 2.2 Subject Eligibility Criteria | 34 |
| 2.2.1 Subject Inclusion Criteria | 34 |
| 2.2.2 Subject Exclusion Criteria | 35 |
| 2.3 Eye-Level Eligibility Criteria | 36 |
| 2.3.1 Eye-Level Inclusion Criteria | 36 |
| 2.3.2 Eye-Level Exclusion Criteria | 37 |
| 2.4 Screening/Baseline Procedures | 37 |
| 2.4.1 Data Collection and Testing | 38 |
| 2.4.1.1 Visual Field Examinations | 39 |
| CHAPTER 3: RANDOMIZATION VISIT | 41 |
| 3.1 Timing | 41 |
| 3.2 Randomization | 41 |
| 3.3 Instructions to Subjects | 41 |
| CHAPTER 4: STUDY TREATMENTS | 42 |
| 4.1 Medical Therapy including Diet | |
| 4.1.1 Acetazolamide | 42 |
| 4.1.1.1 Acquisition | 42 |
| 4.1.1.2 Storage | 42 |
| 4.1.1.3 Accountability of Acetazolamide Supplies | |
| 4.1.1.4 Dosing and Administration | 42 |
| 4.1.1.5 Stopping the Dosage Titration | 43 |
| 4.1.2 Addition of Furosemide | |
| 4.1.3 Assessment of Subject Compliance with Medical Therapy | |
| 4.1.4 Tapering of Medical Therapy | |
| 4.1.5 Discontinuation of Medical Therapy | |
| 4.1.6 Dietary Consultation | 45 |

| 4.2 Optic Nerve Sheath Fenestration | 46 |
|---|---|
| 4.3 CSF Shunting | 46 |
| 4.4 Prohibited Medications, Treatments, and Procedures | 47 |
| 4.5 Concomitant Medications | 47 |
| 4.5.1 Allowed Concomitant Medications | 47 |
| 4.6 Management of the Non-Eligible Eye | 48 |
| 4.7 Treatment during the Treatment Failure Identification Phase | 49 |
| CHAPTER 5: STUDY VISITS AND PROCEDURES | 50 |
| 5.1 Randomized Trial | 50 |
| 5.1.1 Study Visits and Phone Contacts | |
| 5.1.2 Safety Visits | 50 |
| 5.1.3 Study Visit Procedures | 50 |
| 5.1.4 Phone Contact Procedures | 51 |
| 5.1.5 Safety Visit Procedures | 51 |
| 5.2 Treatment Failure Identification Phase | 52 |
| 5.2.1 Follow-up Visits | 52 |
| 5.2.2 Study Visit Procedures | 52 |
| 5.2.3 Phone Contact Procedures | 52 |
| 5.3 Unscheduled Visits | 52 |
| 5.4 Extra Assessments for Subjects Who Appear to be Worsening | 53 |
| 5.5 Early Termination | 53 |
| 5.6 Surgical Malfunction | 53 |
| 5.6.1 Criteria for SMRC Review | 53 |
| 5.6.2 Surgical Malfunction Review by SMRC | 53 |
| 5.6.3 Temporary Treatment Failure | 54 |
| 5.7 Treatment Failure | 54 |
| 5.7.1 Treatment Failure Criteria | 54 |
| 5.7.2 Treatment Failure Review by Adjudication Committee | 54 |
| 5.7.3 Visit Schedule Once Treatment Failure is Reached | 56 |
| CHAPTER 6: TESTING PROCEDURES, QUESTIONNAIRES, CLINICAL ASSESSMENTS, AND | |
| LABORATORY TESTING | |
| 6.1 Testing Procedures | |
| 6.2 Intraocular Pressure | |
| 6.3 Refraction and Visual Acuity | |
| 6.4 Papilledema Grading | |
| 6.5 Perimetry | 57 |

| 6.6 OCT | 57 |
|--------------------------------------------------------------|----|
| 6.7 Lumbar Puncture | 58 |
| 6.8 Quality of Life Assessment | 58 |
| 6.9 Headache Disability Rating | 58 |
| 6.10 Neurologic and Physical Examination | 58 |
| 6.11 Clinical Laboratory Tests | 58 |
| CHAPTER 7: ADVERSE EVENT REPORTING | 59 |
| 7.1 Adverse Events | 59 |
| 7.1.1 Definitions | 59 |
| 7.1.2 Reporting Adverse Events | 59 |
| 7.1.3 Relationship of Adverse Event to Study | 60 |
| 7.1.4 Intensity of Adverse Events | 60 |
| 7.1.5 Coding of Adverse Events | 60 |
| 7.1.6 Outcome of Adverse Event | 61 |
| 7.2 Pregnancy Reporting | 61 |
| 7.3 Timing of Event Reporting | 61 |
| 7.4 Stopping Criteria | 62 |
| 7.4.1 Subject Discontinuation of Study Drug | 62 |
| 7.5 Medical Monitor | 62 |
| 7.6 Independent Safety Oversight | 62 |
| 7.7 Criteria for Suspending or Terminating Overall Study | 62 |
| CHAPTER 8: MISCELLANEOUS CONSIDERATIONS | 63 |
| 8.1 Subject Compensation | 63 |
| 8.2 Subject Withdrawal | 63 |
| 8.3 Confidentiality | 63 |
| CHAPTER 9: STATISTICAL CONSIDERATION | 64 |
| 9.1 Statistical and Analytical Plans | 64 |
| 9.2 Intention-to-Treat Principle | 64 |
| 9.3 Analysis of the Primary Outcome Variable | 64 |
| 9.3.1 Primary Statistical Model | 64 |
| 9.3.2 Adjustment for Baseline Characteristics | 65 |
| 9.3.3 Investigation of Treatment by Covariate Interactions | 65 |
| 9.3.4 Verification of Model Assumptions | 65 |
| 9.3.5 Treatment of Missing Data | 65 |
| 9.4 Analysis of the Secondary Outcome Variables for Efficacy | 66 |

| 9.5 Compliance Outcomes | 67 |
|------------------------------------------------------------|----|
| 9.6 Analysis of Safety and Tolerability Outcomes | 67 |
| 9.6.1 Adverse Events | 67 |
| 9.6.2 Tolerability Outcomes | 68 |
| 9.6.3 Laboratory Test Results and Vital Signs | 68 |
| 9.7 Analysis of Long-Term Follow-Up Data | 68 |
| 9.8 Interim Analyses | 69 |
| 9.8.1 Interim Analyses for Safety | 69 |
| 9.8.2 Interim Analyses for Efficacy | 70 |
| 9.9 Baseline Characteristics | 70 |
| 9.10 Sample Size Determination | 70 |
| CHAPTER 10: DATA COLLECTION AND MONITORING | 73 |
| 10.1 Case Report Forms | 73 |
| 10.2 Study Records Retention | 73 |
| 10.3 Quality Assurance and Monitoring | 73 |
| 10.4 Protocol Deviations | 74 |
| 10.5 Committees and Reading Centers | 74 |
| 10.5.1 Resource Center (RC) | 74 |
| 10.5.2 Visual Field Reading Center (VFRC) | 74 |
| 10.5.3 Photographic Reading Center (PRC) | 75 |
| 10.5.4 Optical Coherence Tomography Reading Center (OCTRC) | 75 |
| 10.5.5 Surgical Quality Assurance Committee (SQAC) | 75 |
| 10.5.6 Surgical Malfunction Review Committee (SMRC) | 75 |
| 10.5.7 Adjudication Committee (AC) | 76 |
| CHAPTER 11: ETHICS/PROTECTION OF HUMAN SUBJECTS | 77 |
| 11.1 Ethical Standard | 77 |
| 11.2 Institutional Review Boards | 77 |
| 11.3 Informed Consent Process | 77 |
| 11.3.1 Consent Procedures and Documentation | 77 |
| 11.3.2 Subject and Data Confidentiality | 77 |
| 11.3.3 Future Use of Stored Specimens | 78 |
| CHAPTED 12. DEEEDENCES | 90 |

### **LIST OF ABBREVIATIONS**

| ABBREVIATION | DEFINITION |
|--------------|---------------------------------------------------------------|
| CC | Coordinating Center |
| CFR | Code of Federal Regulations |
| CRF | Case Report Forms |
| CSF | Cerebrospinal Fluid |
| DSMC | Data Safety Monitoring Committee |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| IIH | Idiopathic Intracranial Hypertension |
| IIHTT | Idiopathic Intracranial Hypertension Treatment Trial |
| ICH | International Conference on Harmonization |
| IND | Investigational New Drug |
| IRB/IEC | Institutional Review Board/Independent Ethics Committee |
| JCHR | Jaeb Center for Health Research |
| MOP | Manual of Procedures |
| MRI | Magnetic Resonance Imaging |
| NEI | National Eye Institute |
| NORDIC | Neuro-Ophthalmology Research Disease Investigator Consortium |
| OCT | Optical Coherence Tomography |
| OCTRC | OCT Reading Center |
| ONSF | Optic Nerve Sheath Fenestration |
| PMD | Perimetric Mean Deviation |
| PRC | Photography Reading Center |
| QoL | Quality Of Life |
| RC | Resource Center |
| RCT | Randomized Clinical Trial |
| SAE | Serious Adverse Experience |
| SIGHT | Surgical Idiopathic Intracranial Hypertension Treatment Trial |
| SMRC | Surgical Malfunction Review Committee |
| SQAC | Surgical Quality Assurance Committee |
| TF | Treatment Failure |
| VFRC | Visual Field Reading Center |
| VPS | Stereotactic Ventriculo-Peritoneal CSF Shunting |

## PROTOCOL SUMMARY

| PARTICIPANT AREA | DESCRIPTION |
|---|---|
| Title | A Multicenter, Partially-Masked, Randomized, Controlled Study of Medical Therapy vs. Medical Therapy plus Optic Nerve Sheath Fenestration vs. Medical Therapy plus Stereotactic Ventriculoperitoneal Cerebrospinal Fluid Shunting in Subjects with Idiopathic Intracranial Hypertension and Moderate to Severe Visual Loss ("SIGHT") |
| Précis | Randomized trial of adults (≥18 years old) with idiopathic intracranial hypertension and moderate to severe visual loss without substantial recent treatment who are randomly assigned to (1) medical therapy, (2) medical therapy plus ONSF, or (3) medical therapy plus VPS. The primary outcome is visual field mean deviation change at first of Month 6 (26 weeks) or time of treatment failure of the eligible eye(s), followed by a continuation study to assess time to treatment failure. The determination of eligible eye(s) is based on meeting the eligibility criteria at baseline. |
| Study Objectives | Primary objective: to determine whether the efficacy of stereotactic ventriculo-peritoneal CSF shunting (VPS) with medical therapy is superior to medical therapy alone or optic nerve sheath fenestration (ONSF) with medical therapy in reducing or reversing visual loss in subjects with idiopathic intracranial hypertension and moderate to severe visual loss. Secondary objective: To assess time to treatment failure over up to 3 years. |
| Study Design | Multi-center randomized single-masked phase 3 clinical trial |
| Study Design | RCT is followed by a treatment failure identification phase (up to 3 years of follow-up total) |
| Number of Sites | ~40 sites |
| Endpoint | Primary Efficacy Outcome: |
| | <ul> <li>Change from baseline to first of Month 6 (Week 26) or time of<br/>treatment failure in PMD (perimetric mean deviation) in eligible<br/>eye(s) with the size V stimulus.</li> </ul> |
| | Key Secondary Efficacy Outcomes: |
| | Time from randomization to treatment failure |
| | CSF pressure measurement by lumbar puncture |
| | Papilledema grade |
| | OCT measures |
| | QOL assessments |
| | <ul> <li>Visual field examination ratings (improved, remained the same, or<br/>worsened)</li> </ul> |
| | Key Safety Outcomes: Vision loss, all reported adverse events |
| | Other Key Outcomes: Change in weight |

| PARTICIPANT AREA | DESCRIPTION |
|---|---|
| Population | Subject Eligibility Criteria |
| - | Inclusion Criteria |
| | 1. Diagnosis of IIH by modified Dandy criteria (Table 4) |
| | 2. Age 18 to <64 years at time of consent |
| | 3. Age 18 to <61 years at time of diagnosis (time of diagnosis is the time at which the patient meets the modified Dandy criteria, usually after the lumbar puncture results are reviewed) |
| | 4. Presence of bilateral papilledema |
| | 5. Lumbar puncture within 6 weeks of screening visit or completed as part of screening: Opening CSF pressure >250 mmH2O or 200 to 250 mmH2O, with at least one of the following: |
| | <ul> <li>Pulse synchronous tinnitus</li> </ul> |
| | Cranial nerve VI palsy |
| | <ul> <li>Echography for disc drusen negative and no other disc<br/>anomalies mimicking disc edema present</li> </ul> |
| | <ul> <li>MRV with lateral sinus collapse/stenosis, partially empty<br/>sella turcica on coronal or sagittal views of MRI, and optic<br/>nerve sheaths with filled out CSF spaces next to the globe on<br/>T2 weighted axial MRI scans</li> </ul> |
| | If the patient was treated with intracranial pressure lowering agents (e.g., acetazolamide) prior to obtaining a lumbar puncture, the agent(s) must be discontinued for at least 24 hours prior to performing the diagnostic lumbar puncture. |
| | 6. At least one eye meeting all eligible eye inclusion criteria and no exclusion criteria. |
| | 7. Able to provide informed consent |
| | 8. Investigator believes participant is a good candidate for the study, including the probability of returning for follow-up. |
| | Exclusion Criteria |
| | 1. Treatment of IIH within the past 3 months with either (1) the maximally tolerated dosage of acetazolamide for at least one week or (2) more than one month of acetazolamide with a cumulative dosage of more than 45 grams |
| | 'Maximally-tolerated dose' is defined as dosage was reached where dosage could not be increased further either because of side effects or because a daily total dosage of 4 grams per day was reached. |
| | If individual discontinued acetazolamide in the past due to side effects individual is only eligible if investigator believes that the individual is likely to tolerate acetazolamide, as it will be prescribed in the study. |
| | 2. Treatment of IIH within the past 3 months with either (1) the maximally tolerated dosage of methazolamide for at least one week or (2) more than one month of methazolamide with a cumulative dosage of more than 4.5 grams |
| | 'Maximally-tolerated dose' is defined as dosage was reached where dosage could not be increased further either because of side effects or because a daily total dosage of 400 mg per day was reached. |
| | 3. Treatment with topiramate within two months and average cumulative dosage for the preceding month of more than 700 mg per week |

| PARTICIPANT AREA | DESCRIPTION |
|---|---|
| | 4. Previous surgery for IIH, including ONSF, CSF shunting, |
| | subtemporal decompression, or venous sinus stenting; gastric surgery for obesity is allowed |
| | 5. Abnormalities on neurologic examination except for papilledema and its related visual loss or cranial nerve VI to VII paresis; <i>if other abnormalities are present, the patient will need to be discussed with the Study Director for study entry.</i> |
| | 6. Abnormal CT or MRI scan (intracranial mass, hydrocephalus, dural sinus thrombus, or arteriovenous malformation) other than findings known to occur with increased intracranial pressure. Abnormalities on MRI that are not known to cause increased intracranial pressure are acceptable. |
| | 7. Abnormal CSF contents: increased cells: > 8 cells; elevated protein: > 45 mg%; low glucose: < 30 mg% (If the lumbar puncture produces a cell count compatible with a traumatic needle insertion, the patient does not need to be excluded if the CSF WBC after correction is 8 cells/mm³ or less - see MOP for calculation. If > 8 cells or > 45 mg% in CSF protein are documented in the CSF or calculated after conversion from a traumatic lumbar puncture, the patient can be discussed with the Study Director for possible inclusion.) |
| | Abnormal blood work-up indicating a medical or systemic condition associated with raised intracranial pressure |
| | 9. Diabetes mellitus with diabetic retinopathy |
| | 10. Ingestion of a drug or substance, or presence of a disorder, that has been associated with increased intracranial pressure within 2 months of diagnosis, such as lithium, vitamin A related products (e.g. Retin-A), or various cyclines (see MOP for conditions and drugs) |
| | 11. Laboratory test results showing severe anemia, leukopenia or thrombocytopenia, renal failure, or hepatic disease, based on the Site Investigator's judgment |
| | 12. Other condition requiring continued use of oral, I.V. or injectable steroids (nasal, inhaled, or topical steroids are allowed since the systemic effects are small). Patients with a condition that resulted in recent or current use of steroids but may be safely tapered off will be handled on a case-by-case basis after discussion with Study Director/co-Director. See MOP for details. |
| | 13. Presence of a medical condition that would contraindicate use of acetazolamide or furosemide or significantly increase surgical risk |
| | 14. Pregnancy or unwillingness for a subject of childbearing potential to use contraception during the first 6 months of the study |
| | Women of childbearing potential must use an acceptable form of birth control. Acceptable forms include oral contraceptives, IUDs transdermal contraceptives, diaphragm, condoms with spermicide, documented surgical sterilization of either the subject or their partner, or abstinence. |
| | 15. Presence of a physical, mental, or social condition likely to affect follow-up (drug addiction, terminal illness, no telephone, homeless) |
| | 16. Anticipation of a move from the site area within six months and unwillingness to return for follow-up at a SIGHT study site |
| | 17. Allergy to pupil dilating drops or narrow angles precluding safe dilation |

| PARTICIPANT AREA | DESCRIPTION |
|---|---|
| | <ul><li>18. Presence of a condition that contraindicates general anesthesia</li><li>19. Participation in an investigational trial within 30 days of enrollment that involved treatment with any systemic drug therapy or therapy that affects the eligible eye(s)</li></ul> |
| | Eye-Level Eligibility Criteria Subjects must have at least one eye meeting all of the inclusion criteria and none of the exclusion criteria. |
| | If both eyes meet eligibility criteria at the baseline examination, both will be included in the primary outcome analysis. |
| | <ul><li>Inclusion</li><li>1. Visual field loss meeting the following criteria based on two full threshold 24-2 size V tests reviewed by the VFRC:</li></ul> |
| | • PMD from -6 dB to -27 dB |
| | <ul> <li>Reproducible visual loss present on automated perimetry<br/>including no more than 15% false positive response</li> </ul> |
| | 2. Visual acuity better than 20/200 (39 or more letters correct) |
| | Exclusion 1. Intraocular pressure currently >28 mm Hg or >30 mm Hg at any time in the past |
| | 2. Refractive error of more than -6.00 or more than + 6.00 sphere or more than 3.00 cylinder with the following exceptions: |
| | • Eyes with more than 6.00 D of myopia of but less than 8.00 D of myopia are eligible if: 1) there are no abnormalities on ophthalmoscopy related to myopia that are associated with visual loss (such as staphyloma, retinal thinning in the posterior pole, or more than mild optic disc tilt), and 2) the individual will wear a contact lens for all perimetry examinations with the appropriate correction. |
| | • Eyes with more than 6.00 D of hyperopia but less than 8.00 D of hyperopia are eligible if: 1) there is an unambiguous characteristic halo of peripapillary edema as opposed to features of a small crowded disc or other hyperopic change related to visual loss determined by the Site Investigator or the PRC Director (or his designate), and 2) the individual will wear a contact lens for all perimetry examinations with the appropriate correction (which can be corrected for perimetry or with the patient's own contact lens with over correction by lens at the perimeter). |
| | Note: Refractive error exclusion and exceptions refer to sphere not spherical equivalent, with cylinder expressed in plus format. |
| | <ol> <li>Other disorders causing visual loss except for refractive error and<br/>amblyopia, including cells in the vitreous or iritis</li> </ol> |
| | 4. Large optic disc drusen on exam or known in previous history (small drusen of the disc can occur with longstanding papilledema and are allowed if not so numerous that investigator determines they are contributing to vision loss) |
| Sample Size | 180 subjects entering randomized trial |
| | • 90% power to detect a difference in mean change of visual field between groups assuming a true population difference between any 2 of 3 groups = 4.5dB with a two-tailed Bonferroni-adjusted significance level of 1.7%, assuming no more than 10% of subjects withdrawing. |

| PARTICIPANT AREA | DESCRIPTION |
|---|---|
| Treatment Groups | Random assignment (1:1:1) to (1) medical therapy, (2) medical therapy plus ONSF, or (3) medical therapy plus VPS. |
| Subject Duration | ~7 months- 3 years |
| Protocol Overview/Synopsis | After signing the informed consent form, potential subjects will be assessed for eligibility, including eliciting medical and neurologic history, measurement of best-corrected visual acuity, visual field testing, ophthalmoscopy with optic disc edema grading, physical examination, and OCT. Questionnaires will be completed. Blood will be drawn for CBC, electrolytes, liver function tests, renal function tests, amylase if not done as part of routine care within 4 weeks and a pregnancy test will be performed (women of childbearing potential). |
| | Two visual field examinations using a size V stimulus will need to be performed at the Screening/Baseline Visit. The size V fields will be sent to the VFRC to confirm eligibility or determine that testing must be repeated for the subject. Eligible individuals will be randomly assigned with equal allocation to |
| | Eligible individuals will be randomly assigned with equal allocation to one of 3 treatment groups: (1) medical therapy, (2) medical therapy plus ONSF, or (3) medical therapy plus VPS. Acetazolamide should be started on the day of randomization. Surgery should be performed as soon as possible, ideally within 3 days of randomization, but not more than 7 days. |
| | Medical therapy will consist of a low sodium weight loss diet and acetazolamide with or without furosemide. Treatment will start with acetazolamide 2 grams per day, with the dose increased as tolerated up to 4 grams per day. If there is no clinical improvement after 2 weeks of maximal dosage of acetazolamide, furosemide will be started at a dose of 40 mg per day (along with potassium) and titrated up to 160-200 mg per day. Pharmacotherapy will be tapered when there is improvement in the papilledema grade, substantial improvement in the PMD and improvement in symptoms or when there is a safety concern. |
| | The primary outcome is measured at the first of 6 months (26 weeks) or time of treatment failure. During the randomized trial, follow-up visits will occur after weeks 4, 8, 16, and 26 (± 7 days). Safety visits will occur after weeks 1 and 2 (± 4 days). Additional office visits may occur as needed. Phone contacts will occur after 12 and 20 weeks (±7 days). |
| | After the 6-month primary outcome visit, subjects will transition to the Treatment Failure Identification Phase for up to 3 years. Ongoing treatment will continue following the guidelines for the first six months as long as treatment failure criteria are not met at which time treatment will be at the discretion of the Site Investigator. Investigators are urged to employ treatments from another arm of the study before other treatments under these circumstances. |

# **Chapter 1: Introduction**

| 2 | 1.1 Background |
|---|---|
| 3 4 | Idiopathic intracranial hypertension (IIH), previously called pseudotumor cerebri, is a disorder of elevated intracranial pressure of unknown cause. Its incidence is rising with the obesity |
| 5<br>6<br>7 | epidemic, with about 22.5 new cases each year per 100,000 overweight women of childbearing age. It affects at least 100,000 Americans. Because of pressure on the optic nerve (papilledema), 86% have visual loss and 10% develop severe visual loss. <sup>1</sup> |
| 8 | We recently completed the Idiopathic Intracranial Hypertension Treatment Trial (IIHTT), a |
| 9 | multicenter, randomized, double-masked, placebo-controlled study of 165 subjects with IIH and |
| 0 | mild visual loss. We showed that the acetazolamide-plus-diet regimen was significantly superior |
| 1 | to placebo-plus-diet for improving perimetric mean deviation (PMD), papilledema grade, quality |
| 2 | of life measures (QoL) and intracranial pressure. <sup>2</sup> |
| 3 | In patients with IIH who have moderate to severe visual loss at presentation, no intervention, |
| 4 | neither medical nor the various surgical treatments, has been verified as efficacious by well- |
| 5 | designed clinical trials. The Neuro-Ophthalmology Research Disease Investigator Consortium |
| 6 | (NORDIC) Network has identified management of moderate to severe visual loss in IIH as an |
| 7 | investigational priority. The NORDIC Executive Committee has provided the guidance for the |
| 8 | development of a second prospective IIH treatment trial, the Surgical IIHTT (SIGHT- |
| 9 | pronounced "Sight"). NORDIC will provide the infrastructure to accomplish the proposed study, |
| 20 | consisting of experienced study leadership, ~40 sites (most of whom had successfully executed |
| 21 | the IIHTT), Coordinating Center, Reading Centers, and an Enrollment Center. The goals of the |
| 22 | proposed study are: (1a) to establish evidence-based treatment strategies to restore and protect |
| 23 | vision in IIH patients with moderate to severe visual loss; (1b) to compare currently used |
| 24 | treatment strategies with respect to the cumulative probability of treatment failure over time to |
| 25 | determine long-term outcomes; (2a) to determine how interventions that purportedly lower |
| 26 | intracranial pressure affect deformation of the peripapillary retinal pigment epithelial – Bruch's |
| 27 | membrane layer (ppRPE/BM layer) using optical coherence tomography (OCT) imaging; and (2b) to determine the predictive value of OCT retinal ganglion cell layer (GCL) thickness at |
| 28<br>29 | baseline for visual outcome. |
| 30 | To address these aims, we will enroll 180 newly diagnosed* IIH patients with a perimetric mean |
| 31 | deviation (PMD) between -6 and -27 dB in at least one eye, as determined by full threshold |
| 32 | standard automated perimetry using the size V stimulus. We will compare the efficacy of 1) |
| 33 | medical therapy alone, 2) surgical intervention via optic nerve sheath fenestration (ONSF) with |
| 34 | medical therapy, and 3) surgical intervention via ventriculo-peritoneal cerebrospinal fluid (CSF) |
| 35 | shunting with medical therapy. Subjects will be followed for an initial 6-month intervention |
| 36 | phase, followed by transition to the treatment failure identification phase with clinical follow-up |
| 37 | at 12 months, 24 months, and 36 months. After one year, there will be quarterly telephone |
| 88 | contact to determine the subject's clinical status. |

SIGHT PROTOCOL V4.0 11Apr2019

1

<sup>\*</sup> Nearly all subjects will be "newly diagnosed;" however, if a patient was previously diagnosed but not treated, they will undergo another evaluation for IIH and visual loss to assess eligibility. We expect this situation to be rare.

| 39 | 1.2 Clinical Experience |
|---|---|
| 40 | 1.2.1 Visual Loss in IIH |
| 41<br>42<br>43<br>44<br>45<br>46<br>47<br>48 | IIH has four stages based on severity of visual loss. The first stage (20% of IIH patients) exhibits papilledema and symptoms, but no visual field loss. The second stage (40% of cases), the target for the IIHTT, is characterized by mild visual field defects and prompts effective intervention. The third stage (30% of cases), a target for the SIGHT, is characterized by moderate visual loss. Stage three patients have symptomatic vision loss and current thinking, without class I or II evidence, suggests that aggressive intervention is required to prevent blindness. In the fourth stage (10% of cases), also a target for the SIGHT, severe visual loss occurs, which can worsen rapidly to blindness. |
| 49<br>50<br>51<br>52<br>53<br>54 | Medical treatments, including diet, acetazolamide, and furosemide, are the interventions usually employed for the first two stages of IIH. Several retrospective studies of obese patients with IIH suggest that weight loss may be associated with reduction in papilledema grade. The IIHTT demonstrated that acetazolamide-plus-diet led to a statistically significant improvement in vision and significant improvements in papilledema grade, CSF pressure, and quality of life measures a 6 months compared to placebo-plus-diet in patients with mild visual loss. |
| 55<br>56 | Surgical treatments, such as ONSF and CSF shunting, with or without medical therapy, are commonly employed in the third and fourth stages of IIH. |
| 57 | 1.2.2 Optic Nerve Sheath Fenestration for IIH |
| 58<br>59<br>60<br>61<br>62 | Hayreh, <sup>3</sup> using a primate model, demonstrated efficacy of ONSF for relief of experimental papilledema. Later, Smith et al. <sup>4</sup> reported successful relief of papilledema in a human after ONSF. ONSF consists of either creating a window or making a series of slits in the optic nerve dural sheath just behind the globe in one eye. This treatment has been used for patients with progressive visual loss, and over 50% of patients with IIH have post-operative headache relief. <sup>5</sup> |
| 63<br>64<br>65<br>66<br>67<br>68<br>69<br>70<br>71<br>72<br>73<br>74<br>75<br>76 | Several hypotheses exist as to the mechanism of action of ONSF. The demonstration of fistula formation <sup>6,7</sup> and some improvement of papilledema in the unoperated eye suggest that ONSF efficacy may be due to local decompression of the subarachnoid space with filtration of CSF into the orbit. CSF pressure may be modestly lowered post-operatively, but the duration and magnitude of this effect is unknown. Another possible long-term mechanism of action of ONSF may be secondary closure of the subarachnoid space via fibrosis at the surgical site, thereby preventing transmission of pressure to the optic nerve head. The success of surgical decompression of the optic nerve, however, may be limited by several factors that are not yet fully understood. Trabeculations within the retrobulbar subarachnoid space may contribute to resistance of bidirectional CSF flow between the optic nerve sheath and the intracranial subarachnoid space; this compartmentalization of CSF, demonstrated in vivo by Killer et al., may be responsible for the occasional failure of the fellow eye to improve after ONSF. On the other hand, there may be free flow from the fenestration site to the full CSF space and a generalized pressure lowering effect may occur. It is not known which if either of these mechanisms prevails. |
| 78<br>79 | A meta-analysis of large case series suggests efficacy of ONSF in IIH. Post-operative visual |

80 reported; however, 13% of patients had worse vision in the post-operative period. A report on 75 eyes from 54 patients undergoing ONSF suggested that patients undergoing ONSF may have 81 substantial long-term failure rates. 12 This study defined perimetric mean deviation worsening as 82 83 > 2 dB deterioration in PMD post-operatively on a single visual field exam. By this criterion, 84 68% of eyes improved or stabilized and 32% worsened. However, these results are suspect since 85 a 2 dB or greater mean deviation worsening is within observed individual retest variability in 86 patients with moderate to severe visual field damage and a confirming visual field should have been required.<sup>13</sup> Although ONSF appears to be helpful in the short term for visual loss, other 87 interventions, such as weight loss or acetazolamide, may have a delayed, but long-term benefit. 88 89 There are no quality of life (QoL) studies of ONSF in IIH. The uncertainties concerning the 90 short- and long-term efficacy and safety of ONSF in moderate to severe IIH can only be 91 addressed with a prospective, randomized, controlled trial.

#### 1.2.3 CSF Shunting for IIH

92

93

94

95

96

97

98

99

100

101 102 Various CSF shunting procedures have been employed for the treatment of IIH, including lumbo-peritoneal (LP), ventriculo-atrial (VA), ventriculo-jugular, and ventriculo-peritoneal (VP) shunting. In general, the indication for a CSF shunting procedure has been failed medical therapy or intractable headache. Most series document efficacy in preserving vision in most cases, but there was a high rate of shunt failure and shunt revisions were often required. While shunting preserved vision in many patients, long-term headache relief was achieved in only 50% over 36 months. Many of the shunts inserted were lumbo-peritoneal; these are now out of favor due to a high complication rate, which includes frequent shunt occlusion, infection, and intracranial hypotension. Stereotactically inserted ventriculo-peritoneal shunts (VPS) have a lower failure and complication rate, and are easier to monitor and adjust.

103 There is no consensus regarding strategies for the rapeutic intervention for IIH patients with 104 moderate to severe visual loss. Furthermore, the mechanisms of action of the treatments and their effectiveness remain uncertain.<sup>23</sup> Various therapies have been used to treat IIH, but prior to the 105 106 IIHTT, their safety and efficacy had not been adequately evaluated in prospective, randomized, 107 controlled trials. Although there are large variations in practice, most physicians wait until there 108 is more advanced visual loss before recommending a surgical intervention. However, all studies 109 evaluating interventions for IIH with more advanced visual loss are anecdotal, retrospective, and 110 uncontrolled. Also, the various surgical procedures for IIH have not been compared with regards to efficacy, safety, complication rate, and long-term outcome. Thus, as confirmed by a recent 111 112 Cochrane review, there is an inadequate evidence base to guide clinicians in management of 113 IIH patients with moderate to severe vision loss. 24

Based on Curry's results and extrapolating to 2014, estimating 2500 CSF shunt surgeries per year at a cost of about \$38,500 per patient, and 250 ONSF surgeries at \$23,000 per patient, surgical costs for IIH are estimated at \$102 million per year. Friesner and colleagues come to a similar conclusion regarding surgical costs. In addition, they estimated in 2007 dollars the total costs due to IIH to be \$444 million per year, so it is imperative that we obtain high quality data regarding the efficacy and safety of surgical treatments for IIH.

#### 1.2.4 Pilot Data for Management of Moderate to Severe Visual Loss in IIH

In 2012, the IIH Study Group performed a retrospective chart review of consecutive newly diagnosed patients that met the modified Dandy criteria for IIH<sup>27</sup> from 30 of the 40 IIHTT sites. All patients were seen between January 2009 and September 2012, and had baseline PMD worse than -8.5 dB in at least one eye, as in the eligibility criteria for the SIGHT; this cutoff was chosen based on equipoise of the IIH Study Group – there was discomfort in randomizing subjects to surgery if they did not have at least -8.5 dB PMD in one eye with size III SITA Standard testing. Patients had undergone medical treatment, ONSF, or CSF shunting. Due to a small number of shunt patients, 3 additional sites were asked to abstract charts. Visual field outcomes (PMD) at 3-12 months after intervention were analyzed. Of 298 subjects meeting eligibility criteria stated above, 91 had pre- and post-intervention Humphrey Field Analyzer data available for analysis. (Table 1).

Table 1. Mean and standard deviation (SD) of the PMD (in dB) of the best eligible eye from each treatment group.

| | Initial | SD | Final | SD | Change | SD |
|---------|---------|-----|-------|-----|--------|-----|
| Medical | -14.6 | 6.2 | -10.2 | 9.2 | 4.4 | 7.4 |
| ONSF | -15.3 | 7.1 | -12.4 | 9.0 | 2.9 | 8.3 |
| Shunt | -17.0 | 6.2 | -8.8 | 8.4 | 8.1 | 7.7 |

Although limited by their retrospective nature, these data suggest that both medical and surgical interventions may be effective for treating IIH patients with moderate to severe visual field loss, and that surgical procedures, especially CSF shunting, may be more effective (Figure 1).



Figure 1. Average PMD in the best eligible eye at initial presentation vs final visit 3-12 months later.

SIGHT PROTOCOL V4.0 11Apr 2019

| 140 | 1.2.5 Use of OCT in Monitoring Papilledema in IIH |
|---|---|
| 141<br>142<br>143<br>144<br>145<br>146<br>147<br>148<br>149 | Papilledema is typically quantified from fundus photographs using the Frisén grading scale. <sup>1</sup> OCT can be used to objectively measure the degree of swelling and monitor treatment effects. Time-domain OCT provides cross sectional images of multiple retinal layers and the peripapillary retinal nerve fiber layer (RNFL) with a resolution of approximately 10 microns. <sup>2-5</sup> OCT has several advantages, based on optics, when compared to photographic imaging. OCT is also reasonably reproducible on repeat measurements in normal eyes and in eyes with glaucoma. <sup>6-11</sup> Limitations include no current algorithm specific for optic disc edema, particularly when it is severe. Fundus photography, the current gold standard and the technique that was used in the IIHTT, requires skilled interpretation of features that can be difficult to quantify. |
| 150<br>151<br>152<br>153<br>154<br>155<br>156<br>157<br>158<br>159<br>160 | Most prior OCT studies have investigated disorders that cause RNFL thinning; few report the effects of papilledema on RNFL or total retinal thickness. Time-domain OCT has been compared to fundus photographs in children with IIH. Another study measured RNFL thickness, using scanning laser polarimetry (SLP) and not OCT, in IIH. OCT has demonstrated subretinal macular fluid in patients with papilledema, we and others have shown RNFL thickening using OCT in patients with acute optic neuritis. He have also found that OCT is superior to SLP in demonstrating and quantifying papilledema. Other studies have compared RNFL thickness in papilledema and pseudopapilledema, but have not compared results with fundus photograph grades. When using time-domain OCT in patients with severe papilledema, there can be inaccurate placement of the peripapillary ring to measure optic disc elevation and RNFL thickness, as well as failure of the algorithm used to measure RNFL thickness. |
| 161<br>162<br>163<br>164<br>165<br>166<br>167 | Newer three-dimensional spectral-domain OCT (SD-OCT) methods, such as the cube scan for data collection, give flexibility to find the exact measures of interest with increased resolution and scanning speed to acquire data over a wider area, thereby reducing sampling errors for higher density and faster scans (512 x 128 axial B-scans for a 6 mm2 area). Coupling these advances with refined algorithms will improve the reproducibility and quantification of papilledema and RNFL alterations, even when swelling obscures the disc borders. Higher scan density should improve measurement of localized RNFL defects, which can be related to visual field loss. |
| 169 | 1.3 Rationale |
| 170 | 1.3.1 Discussion of Study Design |
| 171 | 1.3.1.1 Visual Field Monitoring |
| 172<br>173<br>174<br>175<br>176<br>177 | Patients who are newly diagnosed with IIH with moderate to severe visual field loss (with PMD between -6 dB and -27 dB with full threshold size V testing) may be treated with medical or surgical therapy. The current thinking, without class I or II evidence, suggests that aggressive intervention is required to prevent further visual deterioration and blindness. However, it is unclear if any of these treatments are effective for treating this subset of IIH patients. Patients with milder visual loss may benefit from medical therapy alone, as shown by the IIHTT. |

178 Being an average, the PMD is a summary statistic that is less prone to perimetric variability than 179 using individual or groups of test locations. It is assumed that visual loss by visual field 180 examination best reflects neural damage due to increased intracranial pressure and in the IIHTT 181 correlated well with QoL measures. 182 Standard automated perimetry uses size III stimuli. There is now considerable evidence that 183 automated perimetry using size V stimuli has advantages in patients with moderate to severe visual loss. <sup>29,30,32-36</sup> These advantages include lower retest variability and about one additional 184 log unit (10 dB) of useful dynamic range. Use of the larger size V stimuli also makes for an 185 186 easier test for the patient due to an increase in visual field area in moderate to severely damaged 187 visual fields. In addition, the size V stimulus was recently successfully used in another NEI sponsored clinical trial investigating retinitis pigmentosa.<sup>31</sup> Use in this trial will demonstrate its 188 189 utility for optic neuropathies and we will relate size V results to the conventional size III results. 190 1.3.1.2 OCT Monitoring 191 OCT analysis routines have been developed and optimized for glaucoma. Recent data suggest 192 that OCT appears to be the best imaging modality to monitor papilledema and other optic 193 neuropathies. In the IIHTT OCT sub-study, 89 subjects' (43 acetazolamide and 46 placebo) OCT 194 measurements of swelling, average retinal nerve fiber layer thickness (RNFL), total retina 195 thickness (TRT), and optic nerve head volume (ONHV) were similar in both treatment groups at 196 baseline. At 6 months, the swelling in study eyes was reduced in both groups, but the acetazolamide group showed more reduction in RNFL (174 µm vs. 93 µm, p=0.001), TRT (218 197  $\mu$ m vs. 121  $\mu$ m, p=0.001), and ONHV (4.9  $\mu$ m<sup>3</sup> vs. 2.4  $\mu$ m<sup>3</sup>, p=0.001) when compared with the 198 199 placebo group.<sup>37</sup> 200 Furthermore, OCT showed greater improvements in the optic neural canal shape (inward deviation of the peripapillary RPE/Bruch's membrane borders) in the acetazolamide group than 201 in the placebo group. 38 Sibony et al. 39 in another study showed reduction in the RNFL and less 202 inward deviation of the peripapillary RPE/Bruch's membrane borders following interventions 203

that lower intracranial pressure, such as lumbar puncture, VPS and acetazolamide treatment (see

SIGHT PROTOCOL V4.0 11Apr 2019

204205

Figure 2).



Figure 2. Mean posterior displacement of the RPE-Bruch's membrane complex from pre- to post, following interventions (left to right: LP, VP shunt, ACZ) to lower intracranial pressure in IIH<sup>39</sup>.

We have also shown in a case series that the peripapillary RPE/Bruch's membrane positioning normalized within days of intracranial pressure-lowering procedures. These changes can also be seen in eyes with optic atrophy and no apparent papilledema. The deformation of the RPE/Bruch's membrane position appears to be an acute biomarker of changes in intracranial pressure, whereas the optic nerve morphology (edema) is a chronic biomarker that takes at least 1-2 weeks to respond. In some cases, the RNFL or ONH volume may be decreasing, but the RPE/Bruch's membrane does not change, suggesting that intracranial pressure may not be changing, yet axoplasmic flow may be improving or RNFL loss may be occurring. OCT will be done before lumbar puncture at screening/baseline and again at 6 months, to further characterize RPE/Bruch's membrane changes. The RPE/Bruch's membrane biomarker may represent a non-invasive objective method of monitoring intracranial pressure and, thus, may serve as a surrogate for identifying changes in intracranial pressure.

In another study evaluating 31 IIH patients with visual acuity of 20/25 or worse at presentation, macula ganglion cell layer thickness at presentation was mildly correlated (r=0.44, p=0.005), and at 2-3 weeks after presentation was strongly correlated (r=0.76, p=0.0001), with visual field outcome. Furthermore, a reduction of the ganglion cell layer thickness of > 10  $\mu$ m within 2-3 weeks of presentation was also associated with a worse visual field outcome.

We plan to further study changes in OCT parameters to determine their validity as biomarkers for changes in intracranial pressure and optic nerve damage. Preliminary studies suggest that OCT may facilitate early identification of optic nerve injury due to papilledema and have prognostic significance. We anticipate that OCT will provide information that helps guide treatment decisions.

#### 1.3.1.3 Discussion of Subject Characteristics

This study will enroll 180 individuals with IIH who are 18-63 years of age. This age range represents the population that is most likely to be affected by IIH. Children under 13 will not be included because IIH appears to be a different disease in this age group (no correlation with

235 obesity or gender; often arises from a secondary cause). Adolescents will not be eligible for the SIGHT since attrition in weight loss programs within this group of subjects is substantial, as high 236 as 73% in some reports. 41 Only high intensity behavioral modification targeted towards children, 237 238 combined with physical activity program and/or drug therapies have been shown to be effective 239 in small studies. The SIGHT lacks the expertise and means to safely conduct this therapy of 240 weight management in children. Further, the IIHTT provided data to measure the risk of high 241 dose acetazolamide in adults. No such safety data is known in adolescents and the principal 242 safety measures in the SIGHT will center on preservation of vision and surgical complications. 243 We will exclude pregnant women and prisoners. We anticipate that the cohort will be primarily 244 composed of women in their childbearing years that are overweight. Data available on the prevalence of IIH in the US population is limited. The best information on the demographic 245 246 distribution of this condition comes from the IIHTT. Ninety-eight percent of trial subjects were 247 women with a mean age of  $29 \pm 7.4$  years. With regard to race, 65% of subjects were White, 248 25% were Black, and 10% reported another race. Thirteen percent of IIHTT subjects reported 249 being Hispanic or Latino. As was the case for IIHTT, there will be substantial diversity in the 250 types of enrollment centers used in SIGHT including private and university-based practices in 251 both urban and rural settings. Every effort will be made to enroll a diverse population in the 252 SIGHT.

### 1.3.2 Rationale for Medical and Surgical Treatment

#### 1.3.2.1 Medical Therapy

253

254

255

256257

258

259

260

261

262

263

264

265

266267

Medical therapy will consist of acetazolamide, furosemide when needed, and dietary intervention. The dosage of acetazolamide will be titrated from eight tablets daily (2,000 mg daily) to a maximum of 16 tablets daily (4 gm daily), as tolerated, taken in divided doses (bid) with meals. Four grams daily is the largest dosage used in clinical practice. In the IIHTT, the mean dosage used was 2.5 gm/day; 40% of subjects could tolerate 4 gm/day.

If the subject has side effects that substantially interfere with activities of daily living, we will use the highest dosage of study medication tolerated with a minimum of 1/2 tablet (125 mg acetazolamide) per day. Those failing to clinically improve by two weeks after achieving the maximally tolerated dosage of acetazolamide will be titrated up to 80-100 mg twice daily of furosemide (minimum dosage 20 mg per day) with potassium supplementation of 20 meq for each 40 mg of furosemide, as hypokalemia commonly occurs with this regimen. 42-44 A diet rich in potassium (fresh fruits and vegetables) will be encouraged for those taking furosemide and further supplementation will be given as needed.

All enrolled subjects will be advised to adopt a low sodium weight reduction diet with lifestyle modification developed by the Site Investigator. The treatment plan will be individualized and may include consultation with a dietician or referral to a formal weight loss program. Regression of papilledema and symptoms often occurs with a weight loss of 6% of initial body weight that may take months to achieve. <sup>2,45,46</sup> The IIHTT demonstrated that both the acetazolamide group and the placebo group achieved a reduction in weight. <sup>2</sup> The goal of the intervention in the SIGHT will also be 6% weight loss at six months.

#### 1.3.2.2 Optic Nerve Sheath Fenestration

ONSF consists of either creating a window or making a series of slits in the optic nerve dural sheath just behind the globe. This treatment has been used for patients with progressive visual loss due to IIH. The demonstration of fistula formation<sup>6,7</sup> and some improvement of papilledema in the unoperated eye suggest that ONSF efficacy may be secondary to local decompression of the subarachnoid space with filtration of CSF into the orbit.<sup>8</sup> CSF pressure may be modestly lowered post-operatively, but the duration of this effect is unknown. In a meta-analysis of large case series of ONSF for IIH (Table 2), post-operative visual acuity or visual field results were equal to, or better than, pre-operative vision in 87% of patients reported. However, 13% of patients had worse vision in the post-operative period. Up to 50% of patients have post-operative headache relief with ONSF.<sup>5</sup> A report on 75 eyes of 54 patients undergoing ONSF suggested that patients undergoing ONSF may have substantial long-term failure rates.<sup>12</sup>

Table 2. Case series of visual outcome after ONSF.

| Study | Vision Worse | Vision Not Worse | Total |
|---|---|---|---|
| Hupp <sup>47</sup> | 6 | 11 | 17 |
| Sergott <sup>48</sup> | 0 | 23 | 23 |
| Brourman <sup>49</sup> | 0 | 10 | 10 |
| Goh <sup>50</sup> | 9 | 31 | 40 |
| Corbett <sup>5</sup> | 1 | 21 | 22 |
| Plotnik <sup>51</sup> | 4 | 27 | 31<br>20 |
| Acheson <sup>52</sup> | 3 | 17 | |
| Kelman <sup>53</sup> | 3 | 26 | 29 |
| Banta <sup>54</sup> | 11 | 75 | 86 |
| Yazici <sup>7</sup> | 1 | 16 | 17<br>61<br>50 |
| Alsuhaibani <sup>55</sup> | 2 | 59 | |
| Pineles <sup>56</sup> | 12 | 38 | |
| Fonseca <sup>57</sup> | 3 | 11 | 14 |
| Total: | 13% | 87% | 420 |

#### 1.3.2.3 CSF Shunting

288

289

290

291

292293

294

295

296

297

Various shunting procedures have been employed for the treatment of IIH. In general, the indication for a CSF shunting procedure has been failed medical therapy or intractable headache. The case series document efficacy in preserving vision in most cases (Table 3), but reveal a high rate of shunt failure and, thus, shunt revisions were often needed. Compared to other shunting approaches (e.g., lumbo-peritoneal shunts), stereotactic ventriculo-peritoneal shunts (VPS) have lower failure and complication rates, and are easier to monitor and adjust. While the shunting procedures preserved vision in many patients, long-term headache relief was achieved in only 50% after 36 months in one study.

Table 3. Case series of visual outcome after CSF shunting for IIH (NS = not studied).

| Investigators | Year | Shunt Type | Failures | Vision Worse | Vision Not<br>Worse | Total |
|---|---|---|---|---|---|---|
| Rosenberg <sup>58</sup> 1987 LP/VP/V+ | | 20/37 | 9 | 28 | 37 | |
| Johnston <sup>14</sup> | 1988 | LP/CA/VP/VA | 7/41 | 0 | 36 | 36 |
| Eggenberger <sup>16</sup> | 1988 | LP | 15/27 | 0 | 27 | 27 |
| Shapiro <sup>59</sup> | 1988 | LP | 0/4 | 1 | 3 | 4 |
| Burgett <sup>15</sup> | 1992 | LP | 19/30 | 1 | 29 | 30 |
| Bynke <sup>20</sup> | 1997 | VP | 7/17 | 0 | 17 | 17 |
| Tulipan <sup>60</sup> | 1998 | VP | 0/7 | NS | NS | 7 |
| Maher <sup>61</sup> | 2001 | VP | 3/13 | 0 | 13 | 13 |
| McGirt <sup>19</sup> | 2004 | LP/VP/VA | 23/42 | NS | NS | 42 |
| Abu-Serieh <sup>62</sup> | 2007 | VP 6/9 | | 0 | 9 | 9 |
| Nadkarni <sup>63</sup> | 2008 | LP | 10/40 | NS | NS | 40 |
| Abubaker <sup>21</sup> | 2011 | LP/VP | 12/25 | 0 | 25 | 25 |
| Kandasamy <sup>64</sup> | Kandasamy <sup>64</sup> 2011 VP 5/1 | | 5/17 | 0 | 17 | 17 |
| Sinclair <sup>65</sup> | 2011 | VP/LP | 27/53 | 5 | 48 | 53 |
| Tarnaris <sup>22</sup> | 2011 | LP/VP | 12/29 | 9 | 20 | 29 |
| El-Saadany <sup>66</sup> | 2012 | LP | 8/22 | NS | NS | 22 |
| Yadav <sup>67</sup> | 2012 | LP | 2/24 | 8 | 16 | 24 |
| Huang <sup>68</sup> | 2014 | VP | 7/19 | 1 18 | | 19 |
| Rizzo <sup>69</sup> | 2014 | VP/LP | 4/15 | 0 | 15 | 15 |
| Fonseca <sup>57</sup> | 2014 | VP | 9/19 | 4 | 15 | 19 |
| Total: | | | 40% | 8% | 92% | 374 |

| 298 | 1.4 Study Objectives |
|---|---|
| 299 | 1.4.1 Primary Objective |
| 300<br>301<br>302<br>303<br>304<br>305 | The primary objective is to compare the efficacy of 1) medical therapy, 2) optic nerve sheath fenestration (ONSF) plus medical therapy, and 3) stereotactic ventriculo-peritoneal CSF shunting (VPS) plus medical therapy in newly diagnosed IIH patients with full threshold size V 24-2 PMD between -6 and -27 dB in at least one eye at study entry. Change in the PMD with stimulus size V from baseline to the first of Month 6 or time of treatment failure in the eye(s) qualifying for study entry will be the primary outcome variable. |
| 306 | 1.4.2 Secondary Objectives |
| 307<br>308 | Secondary objectives are to compare changes in the following from baseline to 6 months among the three study groups: |
| 309 | PMD with stimulus size V in the best eye qualifying for study entry |
| 310 | • Papilledema grade (Photographic Reading Center and site investigator ratings) |
| 311 | • OCT measures of: |
| 312 | <ul> <li>Retinal nerve fiber layer thickness</li> </ul> |
| 313 | <ul> <li>Retinal ganglion cell layer thickness</li> </ul> |
| 314 | <ul> <li>Peripapillary retinal pigment epithelial (RPE)/Bruch's membrane deformation</li> </ul> |
| 315 | • CSF pressure |
| 316 | Visual acuity |
| 317<br>318 | <ul> <li>Quality of life (QoL) measures (NEI-VFQ-25 + 10-item neuro-ophthalmic supplement<br/>and the SF-36)</li> </ul> |
| 319 | <ul> <li>Headache disability (HIT-6 Inventory)</li> </ul> |
| 320 | Headache severity |
| 321<br>322<br>323 | Other efficacy outcome variables, determined at Month 6, include treatment failure, surgical failure, presence of headache, presence of transient visual obscurations, and visual field examination ratings (improved, no change, worse) by the Visual Field Reading Center. |
| 324<br>325 | With the exception of CSF pressure, these outcome variables will also be examined at Months 12, 24 and 36. |
| 326<br>327<br>328<br>329 | Of special interest and a very important outcome is the time from randomization to treatment failure. Subjects will be followed for up to 3 years and the number of surgical failures and treatment failures will be analyzed. While a therapy may have a beneficial outcome at 6 months, it may not have a good outcome 1-3 years later; therefore, this is an important analysis. |

| 330 | Measures of safety include the following: |
|---|---|
| 331 | • Adverse events |
| 332 | Serious adverse events |
| 333 | <ul> <li>Procedure complications and transient malfunctions of surgical procedures</li> </ul> |
| 334 | Blood pressure |
| 335<br>336 | • Laboratory test results (CBC with platelet count, electrolytes, potassium, bicarbonate, and liver function tests) |
| 337 | 1.4.3 Other Outcomes |
| 338 | • Anthropometric measures (weight, waist circumference) |
| 339 | 1.5 Potential Risks and Benefits of the Study Interventions |
| 340 | 1.5.1 Known Potential Risks |
| 341 | 1.5.1.1 Visual Loss |
| 342<br>343 | The primary risk of IIH is visual loss associated with papilledema. Subjects reaching treatment failure criteria will remain in the study but will be managed by the site investigators. |
| 344 | 1.5.1.2 Acetazolamide |
| 345<br>346<br>347<br>348<br>349<br>350<br>351<br>352 | Acetazolamide frequently causes paresthesias, altered taste sensation, asymptomatic metabolic acidosis (low serum bicarbonate), and fatigue. There is a small risk of kidney stones, and, very rarely, renal failure from acute tubular necrosis, liver enzyme changes, elevation of serum amylase, blood dyscrasias, Stevens-Johnson syndrome, and aplastic anemia. Based on the IIHTT, we anticipate that renal stones and allergic rashes will occur, though infrequently. Guidance on management of liver enzyme changes and renal stones is provided in the MOP. While there was minimal potassium loss in some IIHTT subjects treated with acetazolamide, there were no instances of hypokalemia requiring potassium supplementation. |
| 353<br>354<br>355<br>356<br>357<br>358<br>359<br>360<br>361 | Subjects will have laboratory studies throughout the study period to monitor their electrolytes. Aplastic anemia can occur in an individual by an idiosyncratic hypersensitivity reaction and cannot be predicted by routine monitoring of the blood count. Some patients may be allergic to acetazolamide, developing a rash (most common reaction), angioedema, stridor, or rarely, anaphylaxis. A history of sulfa allergy will not be an exclusion criterion due to the lack of evidence for cross reactivity with acetazolamide. The study medication will be discontinued immediately if there is any evidence of an allergic reaction. At the conclusion of the subject's participation in the study, their treating physician will arrange a treatment plan independent of the study. |

| 362<br>363<br>364<br>365<br>366<br>367<br>368<br>369<br>370<br>371 | Hypokalemia: Epstein et al. <sup>73</sup> showed no evidence of clinically significant hypokalemia in 92 patients on acetazolamide unless they were also taking other diuretics. We confirmed this in the IIHTT. <sup>2</sup> Since acetazolamide-induced hypokalemia is so uncommon, serum electrolytes will be obtained at 1 month, 4 months, and 6 months (unless subjects develop symptoms of hypokalemia: weakness, fatigue, and muscle cramps). If a subject also requires treatment with furosemide, he/she will have close monitoring of serum electrolytes (including serum sodium and potassium) prior to each change in dosage, to be performed at a local laboratory. The dosage of furosemide will not be increased until it is documented that the potassium level is in the normal range. Once the final furosemide dosage has been reached, electrolytes will be checked a each visit. |
|---|---|
| 372<br>373<br>374<br>375<br>376<br>377 | Aplastic Anemia: Acetazolamide-induced aplastic anemia is dosage independent, usually delayed in onset, and usually fatal. According to prior studies <sup>74,75</sup> , the incidence has been estimated as 1 per 15,000 patient years with a mean age of 71 years (range 56-86 years). The average onset is 3.5 months after initiation of treatment; it rarely occurs after six months of treatment. Monitoring of CBCs is not the standard of care. We will obtain a CBC at baseline and 4 months, and 6 months. |
| 378 | 1.5.1.3 Furosemide |
| 379<br>380<br>381<br>382<br>383<br>384<br>385<br>386<br>387 | Hypokalemia is the most common important side effect of furosemide. Supplemental potassium chloride and, if required, an aldosterone antagonist are helpful in preventing hypokalemia and metabolic alkalosis. Cases of tinnitus and reversible or irreversible hearing impairment and deafness have been reported in people taking furosemide. Reports usually indicate that furosemide ototoxicity is associated with rapid injection, severe renal impairment, the use of higher than recommended doses, hypoproteinemia or concomitant therapy with aminoglycoside antibiotics, ethacrynic acid, or other ototoxic drugs. Excessive diuresis from furosemide can occur that may require measures to prevent dehydration and hypotension. Asymptomatic hyperuricemia can occur and gout may rarely be precipitated. |
| 388<br>389<br>390<br>391 | In summary, common side effects of furosemide are orthostatic hypotension and hypokalemia. Less frequent side effects are hyponatremia, hypocalcemia, hypochloremia, and hypomagnesemia. Also infrequent are cramps, diarrhea, drowsiness, dry mouth, loss of appetite, stomach cramps and photosensitivity. |
| 392 | 1.5.2 Known Potential Benefits |
| 393<br>394<br>395<br>396 | Benefits from participation in the study include assignment to a treatment routinely used in clinical practice, easy access to care for IIH, closer and more careful follow-up assessments evaluating vision. Hopefully, in the future, other people might benefit from this study because of the knowledge that may be gained about IIH. |
| 397 | 1.5.3 Risk Assessment |
| 398 | The risk level is considered to be research involving greater than minimal risk. |

#### 399 **1.6 General Considerations**

The study is being conducted in compliance with the policies described in the study policies document, with the ethical principles that have their origin in the Declaration of Helsinki, with the protocol described herein, and with the standards of Good Clinical Practice (GCP).

Data will be directly collected in electronic case report forms, which will be considered the source data.

### 1.7 Schematic of Study Design



### **Statistical Comparisons**

1° Outcome is Perimetric MD (PMD) change in eligible eye(s) from baseline to first of either 1) Month 6 or 2) time of treatment failure

2° measures at 6 months: Changes in CSF pressure OCT / papilledema changes Changes in quality of life Treatment Failures

### Follow for Remainder of Study for Poor Outcomes

(to find cumulative probability of time to treatment failure in each eligible eye)

406

403 404

405

## 407 **1.8 Schedule of Study Visits and Procedures**

### 1.8.1 Randomized Trial

408

| | | Safety<br>Visit <sup>1</sup> | Safety<br>Visit <sup>1</sup> | | | | | | Primary<br>Outcome |
|---|---|---|---|---|---|---|---|---|---|
| Overview of Study Procedures | SC/BL<br>Visit<br>(-3-0 days) | S Visit<br>1 wk<br>±4 days | S Visit<br>2 wks<br>±4 days | Visit 1<br>4 wks<br>±7 days | Visit 2<br>8 wks<br>±7 days | Phone<br>call<br>12 wks<br>±7 days | Visit 3<br>16 wks<br>±7 days | Phone<br>call<br>20 wks<br>±7 days | Visit 4<br>26 wks<br>±7 days |
| Written Informed Consent | X | | | | | | | | |
| Eligibility Criteria | X | | | | | | | | |
| Med/IIH History/Update | X | | | X | X | | X | | X |
| Physical Exam | X | | | | | | | | |
| Lumbar Puncture | X | | | | | | | | X |
| Questionnaires | X | | | | | | | | X |
| Vital Signs with weight | X | X | X | X | X | | X | | X |
| Ocular Exam | $X^2$ | X | X | X | X | | X | | X |
| Refraction/Acuity | X | X | X | X | X | | X | | X |
| Perimetry | X <sup>3</sup> | X | X | X | X | | X | | $X^3$ |
| Fundus Photographs | X | | X | X | X | | X | | X |
| OCT | X <sup>4</sup> | X | X | X | X | | X | | X <sup>4</sup> |
| CBC with platelet count | X | | | | | | X | | X |
| Metabolic panel w LFTs, amylase and electrolytes | X | | | | | | X | | X |
| Electrolyte testing <sup>5</sup> | | | | X | X | | X | | X |
| Blood sample for storage | X | | | | | | | | |
| Pregnancy test | X | | | | | | | | |
| Adverse Events | X | X | X | X | X | X | X | X | X |
| Concomitant Drug Therapy | X | X | X | X | X | X | X | X | X |
| Randomization | X | | | | | | | | |

SIGHT PROTOCOL V4.0 11Apr2019

PAGE 30 OF 87

| | | Safety<br>Visit <sup>1</sup> | Safety<br>Visit <sup>1</sup> | | | | | | Primary<br>Outcome |
|---|---|---|---|---|---|---|---|---|---|
| Overview of Study Procedures | SC/BL<br>Visit<br>(-3-0 days) | S Visit<br>1 wk<br>±4 days | S Visit<br>2 wks<br>±4 days | Visit 1<br>4 wks<br>±7 days | Visit 2<br>8 wks<br>±7 days | Phone<br>call<br>12 wks<br>±7 days | Visit 3<br>16 wks<br>±7 days | Phone<br>call<br>20 wks<br>±7 days | Visit 4<br>26 wks<br>±7 days |
| Dispense/prescribe acetazolamide | X | | | X | X | | X | | X |
| Prescribe furosemide/potassium as needed | | | | X | X | | X | | X |
| Review Drug Compliance | | X | X | X | X | X | X | X | X |
| Dietary Counseling | X | | | X | X | | X | | X |

Timing of 1 week and 2 week safety visits dependent on treatment group (timing for medical therapy group relative to randomization and timing for surgery groups relative to surgical procedure). The 2 week visit could be skipped if there is marked improvement (see section 5.1.2). One or both safety visits will be repeated after each surgical procedure.

<sup>411 &</sup>lt;sup>2</sup> IOP must be measured at Screening to assess eligibility

<sup>412 &</sup>lt;sup>3</sup>Two sets of FT size V at Screening; same requirement for week 26.

<sup>413 &</sup>lt;sup>4</sup> If LP performed, OCT should be performed prior to LP. Another set of OCT testing after LP is optional at Screening.

For subjects taking furosemide, will be done at local lab prior to each dose increase, once the final dose is reached, and then at each visit

### 415

#### 1.8.2 Treatment Failure Identification Phase

| | | | | Final Study<br>Visit | |
|---|---|---|---|---|---|
| Overview of Study Procedures | Phone Call<br>39 wks<br>±7 days <sup>1</sup> | Visit 5<br>52 wks<br>±7 days | Visit 6<br>104 wks<br>±4 wks | Visit 7<br>156 wks<br>±4 wks | Unscheduled<br>Visit <sup>2</sup> |
| Written Informed Consent | | | | | |
| Eligibility Criteria | | | | | |
| Med/IIH History/Update | | X | X | X | $X^3$ |
| Physical Exam | | | | | $X^3$ |
| Lumbar Puncture | | | | | |
| Questionnaires | | X | X | X | |
| Vital Signs w weight | | X | X | X | $X^3$ |
| Ocular Exam | | X | X | X | $X^3$ |
| Refraction/Acuity | | X | X | X | $X^3$ |
| Perimetry | | X | X | X | $X^3$ |
| Fundus Photographs | | X | X | X | $X^3$ |
| OCT | | X | X | X | $X^3$ |
| CBC with platelet count | | | | | $X^3$ |
| Metabolic panel w LFTs, amylase and electrolytes | | | | | |
| Electrolyte testing <sup>4</sup> | | X | X | X | X |
| Blood sample for storage | | | | | |
| Pregnancy Test | | | | | |
| Adverse Events | X | X | X | X | X |
| Concomitant Drug Therapy | X | X | X | X | X |
| Randomization | | | | | |
| Dispense acetazolamide | | | | | |
| Prescribe furosemide/potassium as needed | | X | X | | X |
| Review Drug Compliance | X | X | X | X | X |
| Dietary Counseling | | X | X | | X |

<sup>416</sup> Telephone contacts will occur quarterly after the year 1 visit

<sup>417</sup> If early termination visit, testing will be the same as the primary outcome visit.

<sup>418 &</sup>lt;sup>3</sup> If clinically indicated

<sup>419 &</sup>lt;sup>4</sup> Only for subjects taking furosemide

Chapter 2: Study Enrollment and Screening/Baseline Testing

#### 421 2.1 Subject Recruitment and Enrollment 422 Study subjects will be recruited from ~40 clinical centers in the United States and Canada. 423 Enrollment will proceed with the goal of 180 subjects entering the randomized trial. A maximum of 400 individuals may be enrolled in the study in order to achieve this goal. Subjects 424 425 who have signed consent and started the screening process may be permitted to continue into the 426 trial, if eligible, even if the randomization goal has been reached. 427 All eligible subjects will be included without regard to gender, race, or ethnicity. There is no 428 restriction on the number of subjects to be enrolled by each site toward the overall recruitment 429 goal. Non-identifying information about individuals who are deemed ineligible or decline to 430 participate in the study will be recorded. 431 Some subjects will have been diagnosed with IIH prior to being referred to the study, whereas 432 others may need to go through the diagnosis and screening process after consent is signed. 433 Neuroimaging studies, diagnostic lumbar puncture, and blood tests are considered routine care 434 regardless of the timing. The patient may have already had a lumbar puncture and blood testing, 435 which may not need to be repeated if performed within 4-6 weeks of enrollment. 436 2.1.1 Informed Consent and Authorization Procedures 437 Potential eligibility may be assessed as part of a routine-care examination. Before completing 438 any procedures or collecting any data that are not part of usual care, written informed consent 439 will be obtained 440 For potential study subjects, the study protocol will be discussed with the potential study subject by study staff. The potential study subject will be given the Informed Consent Form to read. 441 442 Potential study subjects will be encouraged to discuss the study with family members and their 443 personal physicians(s) before deciding whether to participate in the study. 444 A copy of the consent form will be provided to the subject and another copy will be added to the 445 subject's study record. 446 As part of the informed consent process, each subject will be asked to sign an authorization for release of personal information. The investigator, or his or her designee, will review the study-447 specific information that will be collected and to whom that information will be disclosed. 448 449 After speaking with the subject, questions will be answered about the details regarding 450 authorization. 451 A subject is considered enrolled when the informed consent form has been signed.

420

| 452 | | 2.2 Subject Eligibility Criteria |
|---|---|---|
| 453 | | 2.2.1 Subject Inclusion Criteria |
| 454<br>455 | Individual in the | duals must meet all of the following inclusion criteria in order to be eligible to participate study. |
| 456 | 1. | Diagnosis of IIH by modified Dandy criteria (Table 4) |
| 457 | 2. | Age 18 to <64 years at time of consent |
| 458<br>459<br>460 | 3. | Age 18 to <61 years at time of diagnosis (time of diagnosis is the time at which the patient meets the modified Dandy criteria, usually after the lumbar puncture results are reviewed) |
| 461 | 4. | Presence of bilateral papilledema |
| 462<br>463<br>464 | 5. | Lumbar puncture within 6 weeks of screening visit or completed as part of screening: Opening CSF pressure >250 mmH2O or 200 to 250 mmH2O, with at least one of the following: |
| 465 | | a) Pulse synchronous tinnitus |
| 466 | | b) Cranial nerve VI palsy |
| 467<br>468 | | c) Echography for drusen negative and no other disc anomalies mimicking disc edema present |
| 469<br>470<br>471 | | d) MRV with lateral sinus collapse/stenosis, partially empty sella turcica on coronal or sagittal views of MRI, and optic nerve sheaths with filled out CSF spaces next to the globe on T2 weighted axial MRI scans |
| 472<br>473<br>474<br>475 | | If the patient was treated with intracranial pressure lowering agents (e.g., acetazolamide) prior to obtaining a lumbar puncture, the agent(s) must be discontinued for at least 24 hours prior to performing the diagnostic lumbar puncture. |
| 476 | 6. | At least one eye meeting all eligible eye inclusion criteria and no exclusion criteria |
| 477 | 7. | Able to provide informed consent |
| 478<br>479 | 8. | Investigator believes the participant is a good candidate for the study, including the probability of returning for follow-up. |
| 480 | Ta | ble 4. Modified Dandy Criteria for IIH <sup>27</sup> |
| | | 1. Signs and symptoms of increased intracranial pressure |

- 2. Absence of localizing findings on neurologic examination
- 3. Absence of deformity, displacement, or obstruction of the ventricular system and otherwise normal neurodiagnostic studies, except for evidence of increased CSF pressure (>200 mm water). Abnormal neuroimaging except for empty sella turcica, optic nerve sheath with filled out CSF spaces, and smooth-walled non flow-related venous sinus stenosis or collapse, 70 should lead to another diagnosis
- 4. Awake and alert
- 5. No other cause of increased intracranial pressure present

#### 481 2.2.2 Subject Exclusion Criteria

493

494

495

499

500

501

502

503

504

505

506

507

508

509

511

512

513 514

515

516

- 482 Individuals meeting any of the following exclusion criteria at baseline will be excluded from 483 study participation.
- 484 1. Treatment of IIH within the past 3 months with either (1) the maximally tolerated dosage 485 of acetazolamide for at least one week or (2) more than one month of acetazolamide with 486 a cumulative dosage of more than 45 grams
- 487 'Maximally-tolerated dose' is defined as dosage was reached where dosage could not be 488 increased further either because of side effects or because a daily total dosage of 4 grams per day was reached. 489
- 490 If individual discontinued acetazolamide in the past due to side effects, individual is only 491 eligible if investigator believes that the individual is likely to tolerate acetazolamide, as it will be prescribed in the study. 492
  - 2. Treatment of IIH within the past 3 months with either (1) the maximally tolerated dosage of methazolamide for at least one week or (2) more than one month of methazolamide with a cumulative dosage of more than 4.5 grams
- 496 'Maximally-tolerated dose' is defined as dosage was reached where dosage could not be 497 increased further either because of side effects or because a daily total dosage of 400 mg 498 per day was reached.
  - 3. Treatment with topiramate within two months and average cumulative dosage for the preceding month of more than 700 mg per week
  - 4. Previous surgery for IIH, including ONSF, CSF shunting, subtemporal decompression, or venous sinus stenting; gastric surgery for obesity is allowed.
    - 5. Abnormalities on neurologic examination except for papilledema and its related visual loss or cranial nerve VI or VII paresis; if other abnormalities are present, the patient will need to be discussed with the Study Director for study entry.
    - 6. Abnormal CT or MRI scan (intracranial mass, hydrocephalus, dural sinus thrombus, or arteriovenous malformation) other than findings known to occur with increased intracranial pressure. Abnormalities on MRI that are not known to cause increased intracranial pressure are acceptable.
- 510 7. Abnormal CSF contents: increased cells: > 8 cells; elevated protein: > 45 mg%; low glucose: < 30 mg% (If the lumbar puncture produces a cell count compatible with a traumatic needle insertion, the patient does not need to be excluded if the CSF WBC after correction is 8 cells/mm $^3$  or less - see MOP for calculation. If >8 cells or >45mg%in CSF protein are documented in the CSF or calculated after conversion from a traumatic lumbar puncture, the patient can be discussed with the Study Director for possible inclusion.)
- 8. Abnormal blood work-up indicating a medical or systemic condition associated with 517 raised intracranial pressure 518
- 519 9. Diabetes mellitus with diabetic retinopathy

| 520<br>521<br>522 | 10. Ingestion of a drug or substance, or presence of a disorder, that has been associated with increased intracranial pressure within 2 months of diagnosis, such as lithium, vitamin A related products (e.g., Retin-A), or various cyclines (see MOP for conditions and drugs) |
|---|---|
| 523<br>524 | 11. Laboratory test results showing severe anemia, leukopenia or thrombocytopenia, renal failure, or hepatic disease, based on the Site Investigator's judgment |
| 525<br>526<br>527<br>528<br>529 | 12. Other condition requiring continued use of oral, I.V. or injectable steroids (nasal, inhaled, or topical steroids are allowed since the systemic effects are small). Patients with a condition that resulted in recent or current use of steroids but may be safely tapered off will be handled on a case-by-case basis after discussion with Study Director/co-Director. See MOP for details. |
| 530<br>531 | 13. Presence of a medical condition that would contraindicate use of acetazolamide or furosemide or significantly increase surgical risk |
| 532<br>533 | 14. Pregnancy or unwillingness for a subject of childbearing potential to use contraception during the first 6 months of the study |
| 534<br>535<br>536<br>537 | Women of childbearing potential must use an acceptable form of birth control during the first 6 months of the study. Acceptable forms include oral contraceptives, transdermal contraceptives, diaphragm, intrauterine devices, condoms with spermicide, documented surgical sterilization of either the subject or their partner, or abstinence. |
| 538<br>539 | 15. Presence of a physical, mental, or social condition likely to affect follow-up (drug addiction, terminal illness, no telephone, homeless) |
| 540<br>541 | 16. Anticipation of a move from the site area within six months and unwillingness to return for follow-up at a SIGHT study site |
| 542 | 17. Allergy to pupil dilating drops or narrow angles precluding safe dilation |
| 543 | 18. Presence of a condition that contraindicates general anesthesia |
| 544<br>545 | 19. Participation in an investigational trial within 30 days of enrollment that involved treatment with any systemic drug therapy or therapy that affects the eligible eye(s) |
| 546 | 2.3 Eye-Level Eligibility Criteria |
| 547<br>548 | To be eligible, an individual must have at least one eye meeting the following inclusion criteria and none of the exclusion criteria. |
| 549 | If both eyes meet eligibility criteria, then both will be included in the primary outcome analysis. |
| 550 | 2.3.1 Eye-Level Inclusion Criteria |
| 551<br>552 | 1. Visual field loss meeting the following criteria based on two full threshold 24-2 size V tests reviewed by the VFRC: |
| 553 | PMD from -6 dB to -27 dB |
| 554<br>555 | <ul> <li>Reproducible visual loss present on automated perimetry including no more than 15% false positives</li> </ul> |
| 556 | 2. Visual acuity better than 20/200 (39 or more letters correct) |
# **2.3.2** Eye-Level Exclusion Criteria

- 1. Intraocular pressure currently >28 mm Hg or >30 mm Hg at any time in the past
- 2. Refractive error of more than -6.00 or more than +6.00 sphere or more than 3.00 cylinder with the following exceptions:
  - Eyes with more than 6.00 D of myopia but less than 8.00 D of myopia are eligible if:
    - 1. there are no abnormalities on ophthalmoscopy or fundus photos related to myopia that are associated with visual loss (such as staphyloma, retinal thinning in the posterior pole, or more than mild optic disc tilt), and
    - 2. the individual will wear a contact lens for all perimetry examinations with the appropriate correction.
  - Eyes with more than 6.00 D of hyperopia but less than 8.00 D of hyperopia are eligible if:
    - 1. there is an unambiguous characteristic halo of peripapillary edema as opposed to features of a small crowded disc or other hyperopic change related to visual loss determined by the Site Investigator or the PRC Director (or his designate), and
    - 2. the individual will wear a contact lens for all perimetry examinations with the appropriate correction (which can be corrected for perimetry or the patient's own contact lens with over correction by lens at the perimeter).

Note: Refractive error exclusion and exceptions refer to sphere not spherical equivalent, with cylinder expressed in plus format.

- 3. Other disorders causing visual loss except for refractive error and amblyopia, including cells in the vitreous or iritis
- 4. Large optic disc drusen on exam or in previous history (small drusen of the disc can occur with longstanding papilledema and are allowed if not so numerous that investigator determines they are contributing to vision loss)

### 2.4 Screening/Baseline Procedures

After informed consent has been signed, a potential subject will be evaluated for study eligibility through the elicitation of a medical history, performance of an ophthalmic exam including visual acuity testing and visual field testing, physical examination by study personnel and local laboratory testing if needed to screen for exclusionary medical conditions.

- Screening/baseline assessments must be completed within 3 days of signing the consent form.
- The only exceptions are 1) if there are perimetry performance issues requiring repeat examinations; 2) if there are unforeseen circumstances that delay the evaluation such as transportation issues, weather related delays or work-related issues. If an exception occurs, two additional days are allowed. During the screening/baseline visit, especially if there are unforeseen delays, the Site Investigator has the option to begin acetazolamide using the titration schedule in section 4.1.1.4.

| 595<br>596 | Individuals who do not initially meet study eligibility requirements may be rescreened at a later date per investigator discretion. |
|---|---|
| 597<br>598<br>599 | Individuals who meet study eligibility requirements and agree to participate must discontinue any medications being used to treat IIH, except for acetazolamide. All diuretics other than acetazolamide must be discontinued immediately. |
| 600 | 2.4.1 Data Collection and Testing |
| 601 | The following procedures will be performed/data collected/eligibility criteria assessed: |
| 602 | <ul> <li>Inclusion and exclusion criteria assessed</li> </ul> |
| 603 | <ul> <li>Demographics (date of birth, sex, race and ethnicity)</li> </ul> |
| 604 | Contact information |
| 605 | Medical history |
| 606 | Concomitant medications |
| 607 | QoL questionnaires |
| 608 | HIT-6 questionnaire |
| 609 | Physical examination to include: |
| 610<br>611 | <ul> <li>Weight, height, waist circumference, vital signs including measurement of blood<br/>pressure and pulse</li> </ul> |
| 612 | <ul> <li>Neurologic exam</li> </ul> |
| 613 | • Refraction |
| 614 | <ul> <li>Visual Acuity tested following refraction using ETDRS charts</li> </ul> |
| 615 | <ul> <li>Humphrey Visual Field testing (see section 2.4.1.1 below)</li> </ul> |
| 616 | • Intraocular Pressure (Goldmann tonometry) |
| 617 | <ul> <li>Ophthalmoscopy with optic disc edema grading (Frisén scale)</li> </ul> |
| 618 | <ul> <li>Biomicroscopy</li> </ul> |
| 619 | <ul> <li>Fundus photographs</li> </ul> |
| 620 | <ul> <li>Optical Coherence Tomography (OCT)* (optic nerve head and macula)</li> </ul> |
| 621<br>622 | • Blood testing (CBC, electrolytes, liver function tests, renal function tests, amylase) if not done as part of routine care within 4 weeks (to be used in screening) |
| 623<br>624 | <ul> <li>Urine or serum pregnancy test for all women who have reached menarche and are<br/>premenopausal and are not surgically sterile</li> </ul> |
| 625<br>626 | • Blood draw for storage (at screening only, with subject approval, discarded if patient not enrolled): |

- With subject agreement, up to 20 ml of blood may be drawn and stored to use in future research of IIH.
- Lumbar puncture (if not completed within 6 weeks of screening visit)
- \*If lumbar puncture done as part of screening, OCT testing should be done *before* the lumbar puncture. Another set of OCT testing *after* the lumbar puncture is optional.

#### 2.4.1.1 Visual Field Examinations

632

639

640

641642

643

644 645

646

647

648

- At the screening visit, a Humphrey visual field result with 24-2 SITA-standard program using stimulus size III may be performed prior to two size V tests if a recent size III result is not available. The size III test can be used as a guide as to whether the subject is likely to have at least one eye meet eligibility criteria when size V testing is done.
- PMD using the size III stimulus should be approximately in range of -8.5 to -30 dB.
- Two size V stimulus fields will be performed in each eye.
  - The two size V stimulus visual field examinations will be transmitted to the Visual Field Reading Center which will evaluate the visual field results: In order for an eye to qualify for the trial, the average PMD with stimulus size V will have to be equal to or worse than -6 dB and better than -27 dB.
  - If the Visual Field Reading Center confirms that the subject is eligible for randomization, it will document the average mean deviation of the two size V tests as well as which eyes qualify as eligible eyes.
  - If the Visual Field Reading Center finds performance issues on the perimetry results, the examination will need to be repeated for the subject to be considered for the randomized trial.
- 649 Depending on the subject's condition (e.g., suspected visual deterioration, fatigue), perimetry
- 650 may be repeated later that day, or up to the 3-day deadline for randomization; the only exception
- being if a perimetry result is unreliable and requires a repeat examination, the site will have an
- additional two working days to complete the visual field examination. These additional sets of
- 653 perimetry examinations will be submitted to the Visual Field Reading Center for
- 654 confirmation/denial of eligibility.
- There will be times that perimetry results are not reliable and a repeat examination will be
- 656 necessary. This may occur not only at the screening/baseline visit but also at any visit. Whenever
- 657 two examinations are required (baseline, 6 months, treatment failure protocol) the following
- outcomes are possible:
- 1. Two examinations performed and: (1) performance criteria are met and (2) pathophysiologic appropriate visual field patterns match. The average of the mean deviations is used for the outcome. Acceptable performance criteria are: the false positive rate is less than 15%, the false negative rate is judged not to be excessive for the amount of visual loss, and gaze tracking data confirms acceptable fixation. All data from eyes in the study must meet these criteria; only results from eyes that do not meet these criteria

| 565<br>566 | | 1 | retested. |
|---|---|---|---|
| 667<br>668 | 2. | | conditions listed in 1 are not met, for a particular eye (or eyes), then for that eye (or the following should be done: |
| 669<br>670 | | a. | a 3 <sup>rd</sup> examination will be performed; if 2 of the examinations meet VFRC criteria, these 2 will be averaged for the outcome |
| 671<br>672<br>673<br>674 | | b. | if 2 of the 3 examinations <u>do not</u> meet VFRC performance standards, the VFRC will discuss the subject's performance with the Site Perimetrist (masked) to determine the reason for poor results, assessing drowsiness, headache, effort and lens alignment |
| 675<br>676<br>677 | | c. | if any of the above issues can be remedied, further visual field examinations will be performed under the new conditions until 2 acceptable tests are completed; the PMD average of these two twill be used for analysis |
| 678 | | d. | if no reliable results are obtainable, the data will be treated as a missing value |

| 679 | Chapter 3: Randomization Visit |
|---|---|
| 680 | 3.1 Timing |
| 681<br>682 | Randomization should occur within 3 days of the start of screening/baseline testing, once the patient has met criteria for eligibility. |
| 683 | 3.2 Randomization |
| 684<br>685 | Prior to randomization, the subject's understanding of the study protocol and willingness to participate and accept assignment to any of the three treatment groups should be confirmed. |
| 686<br>687 | Randomization will occur on the study website after eligibility is verified and the VFRC has approved randomization of the subject. |
| 688<br>689<br>690<br>691 | Once a study subject is randomized, that subject will be counted regardless of whether the assigned treatment is received. Thus, the investigator must not proceed to randomize an individual until he/she is convinced that the individual is eligible and will accept whichever treatment group is assigned through randomization. |
| 692 | Subjects will be randomly assigned with equal allocation to one of the three treatment groups. |
| 693 | medical therapy |
| 694 | medical therapy plus ONSF |
| 695 | medical therapy plus VPS |
| 696<br>697<br>698 | Using a permuted block design, randomization will be stratified by PMD (average of 2 size V stimulus tests) in the eligible eye(s) (-6 dB to >-12 dB; -12 dB to >-20 dB; -20 dB to -27 dB). If a subject has two eligible eyes, the average PMD of the two eyes will be used for stratification. |
| 699 | 3.3 Instructions to Subjects |
| 700<br>701<br>702<br>703<br>704 | Subjects in all groups will be dispensed acetazolamide (see section 4.1) and receive dietary counseling (see section 4.1.6). Acetazolamide should be started on the day of randomization unless the Site Investigator deems delays occurring during the screening/baseline examination may be harmful to the patient. In this case, the acetazolamide titration according to section 4.1.1.4 may be started prior to randomization. |
| 705<br>706 | For subjects in the two surgery groups, surgery should be performed as soon as possible, ideally within 3 days of randomization, but not more than 7 days |

# **Chapter 4: Study Treatments**

# 4.1 Medical Therapy including Diet

#### 4.1.1 Acetazolamide

### 4.1.1.1 Acquisition

707

708

709

710

711

712

713

714715

716

718

719

720

721

722 723

724

Taro Pharmaceutical Industries will supply commercially available 250 mg acetazolamide tablets in bottles of 100. Supplies will be shipped to the study central pharmacy, which will package, label, and distribute the drug kits to the sites. Sites will dispense acetazolamide at visits during the 6-month randomized trial. At the 6-month visit, the subject will be given a prescription for acetazolamide and it will be the subject's responsibility to obtain the drug.

**Table 5. Composition of Acetazolamide** 

| Component and Quality Standard | F | Strength | |
|---------------------------------|-------------|-----------|-------|
| (and Grade, if Applicable) | Function | mg/tablet | % |
| Acetazolamide, USP | Active drug | 250.0 | 48.56 |
| Lactose NF Monohydrate 200 mesh | | 200.0 | 38.85 |
| Corn Starch NF/EP | | 48.0 | 9.32 |
| Gelatin NF | | 3.2 | 0.62 |
| Glycerine USP | | 1.6 | 0.31 |
| Purified Water USP/EP (1) | N/A | (80.00) | |
| Talc USP | | 9.0 | 1.75 |
| Sodium Starch Glycolate NF/EP | Binder | 1.5 | 0.29 |
| Magnesium Stearate NF/EP | Lubricant | 1.5 | 0.29 |
| Total | | 514.8 | 100 |

### 717 **4.1.1.2 Storage**

All study-supplied medication must be kept in a secure, safe area under recommended storage conditions as stated on the labeling with access limited to persons directly involved in the study.

### 4.1.1.3 Accountability of Acetazolamide Supplies

The site must maintain accurate records (including dates) of receipt, dispensing, return, and destruction of the study acetazolamide. Further details on the drug accountability process will be described in the manual of procedures.

#### 4.1.1.4 Dosing and Administration

- All subjects in the three groups will be given acetazolamide with instructions for use.
- The study will use 250 mg tablets of acetazolamide.
- Tablets will be divided into two doses, taken with meals.

- The initial dose will be 1,000 mg twice day and then increased.
- Beginning on Day 3, the dose will be increased by 250 mg every 2 days until a dosage of 4
- grams daily (16 tablets) is reached (day 17) or adverse events (including side effects that
- interfere with activities of daily living) prohibit increasing the dosage further.
- During the titration period, subjects will be instructed to call the Site Coordinator to report any
- intolerable adverse events. The subject may need to be seen for an unscheduled visit for clinical
- assessment.

735

Table 6. Acetazolamide titration schedule (number of 250 mg tablets)

| Start Day | End Day | Breakfast | Dinner | Total Daily |
|-----------|---------|-----------|--------|--------------|
| 1 | 2 | 4 | 4 | 8 (2000 mg) |
| 3 | 4 | 4 | 5 | 9 (2250mg) |
| 5 | 6 | 5 | 5 | 10 (2500 mg) |
| 7 | 8 | 5 | 6 | 11 (2750 mg) |
| 9 | 10 | 6 | 6 | 12 (3000 mg) |
| 11 | 12 | 6 | 7 | 13 (3250 mg) |
| 13 | 14 | 7 | 7 | 14 (3500 mg) |
| 15 | 16 | 7 | 8 | 15 (3750 mg) |
| 17 | | 8 | 8 | 16 (4000 mg) |

736

- 737 If the subject is unable to tolerate the initial acetazolamide dosage, the dosage may be lowered to
- 738 3 tablets daily. The dosage may be subsequently decreased by one tablet every other day (or
- sooner if the subject is substantially symptomatic) if the subject is unable to tolerate it. If the
- subject is then able to tolerate the lower dosage, the daily dosage should be increased according
- to the table above, or more slowly at the Site Investigator's discretion. Additional attempts to
- increase the acetazolamide dosage beyond 17 days may be initiated at the Site Investigator's
- discretion, but not above a total of 4 grams per day. The dosing level achieved by Day 90 will be
- considered the subject's final dosage. This dosage will be maintained through the remainder of
- the treatment period unless the subject improves such that the dosage can be tapered or develops
- 746 intolerable side effects.
- 747 If the acetazolamide is not tolerated at a dosage of 250 mg, then 125 mg (1/2 tablet) will be tried.
- 748 If this is not tolerated, furosemide will be initiated as described in section 4.1.2.

# 749

### **4.1.1.5** Stopping the Dosage Titration

- 750 The Site Investigator can stop or decrease the dosage titration if the subject has reached maximal
- benefit (in the SI's opinion) or there is a safety concern. He/she can consult the Study co-
- 752 Director as necessary.
- 753 See section 4.1.4 below for tapering details regarding VPS group.

# **4.1.2** Addition of Furosemide

If a participant cannot tolerate any dose of acetazolamide or fails to improve clinically (for example, worsening on the basis of: 1) subject report of progressive visual loss, 2) papilledema is worsening, 3) OCT measures are worsening, 4) ETDRS acuity worsens more than 4 letters, or 5) PMD worsens more than 2 dB) after 2 weeks on the maximally tolerated dosage of acetazolamide, furosemide will be added, initiated at 20 mg bid. If the decision is unclear, the case should be discussed with the Study co-Director.

The furosemide dose will be increased up to a maximum of 80 mg bid unless adverse events prohibit further dosage increase, with electrolytes checked ~4 days after each dose increase. After ~4 days of furosemide treatment, electrolytes will be checked (including serum sodium and potassium). If sodium and potassium are normal, the dose will be increased to 40 mg bid. Again after ~4 days, electrolytes will be checked and if normal the dose will again be increased to 60 mg bid and then if after another ~4 days and normal sodium and potassium, the dose will be increased to 80 mg bid and electrolytes checked after ~4 days. Subsequently, electrolytes will be checked at every visit as long as furosemide is being taken. Standard of care electrolyte testing will be done at a local laboratory.

- An unscheduled visit may be needed to initiate furosemide.
- Subjects requiring furosemide will be given a prescription for the medication (the study will not provide the drug). 20 meq of potassium per day will be prescribed to take concomitant with furosemide and increased by 20 meq per day for each 40 mg of furosemide dosed.
- If the Site Investigator determines there has been improvement with a dose of 80 mg bid (160 mg/day) and expects that a higher dosage may be beneficial, the dose may be increased to 100 mg bid (200 mg/day) with close monitoring for hypokalemia and hyponatremia.

Table 7. Furosemide titration schedule (20 or 40 mg tablets may be dispensed)

| Start Day | End Day | Breakfast | Dinner | Total Daily<br>(20 mg) |
|-----------|---------|-----------|--------|------------------------|
| 1 | 2 | 1 | 1 | 2 (40 mg) |
| 4 | 5 | 2 | 2 | 4 (80 mg) |
| 8 | 9 | 3 | 3 | 6 (120 mg) |
| 12 | 13 | 4 | 4 | 8 (160 mg) |
| *16 | 17 | 5 | 5 | 10 (200 mg) |

\*This optional dosage escalation is continued to 200 mg per day only if the Site Investigator determines there has been improvement up to this point and expects that a higher dosage may be beneficial, with close monitoring for hypokalemia and hyponatremia.

### 4.1.3 Assessment of Subject Compliance with Medical Therapy

Subjects will be asked to bring the used study drug bottles to each visit. At each study visit during the first 6 months, the subject's compliance with the acetazolamide dose will be assessed

| 786<br>787 | by pill counts and chloride levels. If the chloride level is not below normal limits, whether the subject is taking the drug should be questioned unless he/she was prescribed a very low dosage. |
|---|---|
| 788 | 4.1.4 Tapering of Medical Therapy |
| 789<br>790<br>791<br>792<br>793 | All subjects will have their pharmacotherapy tapered when the Site Investigator believes that the dosage should be decreased if he/she believes the subject has achieved maximal benefit. For example if the papilledema grade becomes < 1 in both eyes, and the PMD has improved substantially and IIH symptoms are not interfering with activities of daily living, the taper could begin. |
| 794 | The Site Investigator can also taper pharmacotherapy when subject safety dictates a change. |
| 795<br>796 | For subjects in the VPS group, the acetazolamide dosage should be tapered starting on the day of the surgery. See the MOP for details. |
| 797<br>798<br>799 | Otherwise, it is suggested that dosages of each drug be tapered in increments of 25% of the maximum daily dose of one or both study drugs biweekly until either the patient is off medications or reaches a dosage where there is recurrence or worsening of IIH. |
| 800<br>801 | The Site Investigator may consult with the Study co-Director at any time regarding tapering if needed. |
| 802 | 4.1.5 Discontinuation of Medical Therapy |
| 803<br>804<br>805 | Subjects who permanently discontinue taking study medication should be encouraged to remain in the study off medication and continue to be seen according to their original study visit schedule, but will not have routine blood testing performed. |
| 806 | Discontinuation of therapy will be reported on either a visit or phone contact form. |
| 807 | 4.1.6 Dietary Consultation |
| 808<br>809<br>810 | All subjects will be advised to adopt a low sodium weight reduction diet with lifestyle modification by the Site Investigator. The treatment plan will be individualized and may include consultation with a dietician or referral to a formal weight loss program. |
| 811 | |

# **4.2 Optic Nerve Sheath Fenestration**

- ONSF will be performed by a qualified orbital surgeon, with timing indicated below. See MOP for orbital surgeon qualifications. Either a medial or supero-medial lid crease approach may be utilized (see MOP more details). The surgery will make a window in the dural sheath of at least 4 mm in length under the operating microscope. The procedure will be considered successful if CSF egress is noted at the time of fenestration. Post-operative visits will be performed according to the surgeon's usual routine.
  - If both eyes meet study entry criteria, ONSF will be performed on the eye with the worst PMD first, ideally within three days of randomization. If the other eye still meets eye-level eligibility criteria at two weeks after surgery on the first eye, ONSF will be performed on the second eye. If the second eye improves at two weeks after surgery on the first eye and no longer meets eligibility criteria, ONSF will not be performed on that eye.
  - If only one eye meets entry criteria as an eligible eye, ONSF will be performed on the eligible eye ideally within three days of randomization.
    - If the second eye is not eligible for the study because visual field MD is too good, but the eye worsens (i.e. PMD -6 dB or worse with size V perimetry at any time during study follow-up), ONSF will be performed on the non-eligible eye. Also, if the non-eligible eye meets criteria for temporary treatment failure (see section 5.6.3 below), it will be operated on even if the PMD is not worse than -6 dB.
    - If the second eye is not eligible for the study because visual loss is too severe, ONSF will be considered at two weeks after surgery on the eligible eye.

See section 4.6, Management of the Non-Eligible Eye, for exceptions.

Administration of intravenous and topical corticosteroids is permitted intra-operatively, but systemic corticosteroids are not to be administered post-operatively (see MOP for details). Medical therapy will be continued until the Site Investigator believes that the dosage should be stopped or decreased because the subject has improved; he/she may contact the Study co-Director to decide on how to proceed. See section 4.1.4, Tapering of Medical Therapy.

### 4.3 CSF Shunting

CSF shunt surgery will occur ideally within 3 days of randomization by a certified neurosurgeon. See MOP for surgeon qualifications. Using a frameless image-guided stereotactic system, a ventricular shunt catheter will be positioned in the lateral ventricle of the cerebral hemisphere not associated with speech. The ventricular catheter will be connected to an adjustable valve and the distal shunt system will be placed in the peritoneal cavity. Post-operative computed tomography of the brain will be obtained to confirm shunt tip placement. Post-operative visits will be performed according to the surgeon's usual routine.

- Since the purpose of this procedure is to normalize CSF pressure, the Site Investigator will taper medical therapy at the time of the surgery and then further if/when he/she is confident that the
- VPS is working (see section 4.1.4, Tapering of Medical Therapy).

# 4.4 Prohibited Medications, Treatments, and Procedures

854 Corticosteroids, topiramate, methazolamide, and additional diuretics (other than furosemide)

may not be used during the study period (except intra-operative corticosteroids with ONSF).

Should a subject begin an excluded treatment during the trial, this will be reported on a visit or

phone contact form. The Study Director/co-Director will determine whether there is a potential

safety risk and whether study treatment needs to be discontinued.

857

859

860

861

862

863

864

865

866

867

868869

870

871872

873

874

875

876

877

878

882

883

884

Other treatments for IIH, including bariatric surgery and transverse sinus stenting, will not be allowed during the first six months.

#### 4.5 Concomitant Medications

#### 4.5.1 Allowed Concomitant Medications

All concomitant medications must be used in accordance with approved labeling and as prescribed unless they are commonly used off-label for the prescribed purpose.

Headaches may persist as a major management problem in IIH patients after study treatments have been given. R2,83 The headache can be treated with standard prophylactic vascular headache remedies: non-steroidal anti-inflammatory drugs and tricyclic antidepressants may be effective. Low dosage amitriptyline is suggested; the initial dosage will be 10 mg at bedtime, gradually increasing to a maximum of 50 mg at bedtime, if needed. Weight gain is a well-known side effect of amitriptyline; by using a low dosage and monitoring the subject's weight, we anticipate minimizing this untoward effect. Acute headache may be treated with non-steroidal anti-inflammatory drugs (naproxen 500 mg bid), but their use will be limited to no more than three days per week to prevent analgesic rebound (medication overuse) headache. Table 8 below gives the Site Investigator a group of medications from which to choose. These medications should not be used more than 3 days per week.

Table 8. Medications available for the symptomatic treatment of headache.

| Medication* | Maximum Daily Dosage** |
|-----------------------------------|------------------------|
| Naproxen sodium | 1 gram |
| Acetaminophen | 1500 mg |
| Aspirin | 1950 mg |
| Ibuprofen | 1600 mg |
| Acetaminophen with codeine 30 mg | 4 tablets |
| Butalbital/APAP or Butalbital/ASA | 4 tablets |

<sup>\*</sup> Acetaminophen, aspirin, and non-steroidal anti-inflammatory drugs are preferred.

There is no single agent that will be effective and tolerated by all subjects needing prophylactic headache therapy. Table 9 below takes into consideration the undesirable side effects of many available agents for headache prevention. Gabapentin has few drug interactions, but may

<sup>\*\*</sup> Symptomatic treatment should be limited to 3 times weekly or less to prevent analgesic rebound (medication overuse) headache. Subjects requiring symptomatic headache treatment more than 3 times per week should be prescribed a preventive medication.

increase the serum concentration of barbiturates and morphine. The selective serotonin reuptake inhibitors may produce a small amount of weight gain within the first year of usage. Protriptyline is the least sedating of the tricyclic antidepressants and is least likely to produce weight gain of medications in this class, but also may not be as effective at headache relief.

Table 9. Preventive medications for headache.

| 1 <sup>st</sup> -Tier Medications | |
|---|---|
| Medication | Suggested Starting and Final Dosages |
| Amitriptyline | 10 mg qhs, up to 50 mg qhs if needed* |
| Vivactil <sup>™</sup> (protriptyline) | 5 mg qhs, up to 10 mg bid if needed* |
| Naproxen | Up to 1 gram daily in divided doses |
| Nortriptyline | 25 mg qhs |
| * May be associated with weight gain; monitoring required | |
| 2 <sup>nd</sup> -Tier Medications | |
| Medication | Suggested Starting and Final Dosages |
| Gabapentin | 100 mg qhs, up to 400 mg TID if needed |
| Fluoxetine | 20 mg daily |

Subjects already taking preventive medication for headache at study entry may continue using their preventive medication *unless they are taking topiramate*. It is uncertain if the carbonic anhydrase inhibition associated with topiramate is sufficient to have potential therapeutic value in IIH; this could confound the results of the study.

### 4.6 Management of the Non-Eligible Eye

In general, non-eligible eyes are treated the same as eligible eyes. The non-eligible eye will have the same evaluations as the eligible eye. The only difference between eligible and non-eligible eyes is only the eyes that qualify at baseline (i.e., eligible eyes) will be included in the primary outcome analysis.

If a non-eligible eye worsens, the protocol for worsening of an eligible eye will be used. In the case of medical therapy, the dosage protocols for acetazolamide and if needed furosemide will be used. If there is worsening of a non-eligible eye in the optic nerve sheath fenestration group, the procedure will be performed on the 2<sup>nd</sup> eye if PMD worsens to -6 dB or worse with size V perimetry at any time during study follow-up or if the non-eligible eye meets criteria for temporary treatment failure (see section 5.6.3 below). If there is worsening of a non-eligible eye in the CSF shunting arm, medical therapy will be given and an evaluation for shunt failure will be done. Non-eligible eyes can be used to classify the subject as a treatment failure.

If only one eye meets study entry criteria and the other eye has worse vision by PMD than the eligible eye (e.g. PMD worse than -27 dB, refractive error too great, previous damage to the eye due to trauma, inflammation or infection) treatment of the eligible eye will take precedence; so in the case of optic nerve sheath fenestration, the eligible eye will be done first. However, there may be situations where the non-eligible eye requires the first operation. For example, if fixation is threatened only in the non-eligible eye. If the Site Investigator has concerns about the non-

| 913<br>914 | eligible eye and believes it should be operated first, a decision will be made with the Study co-<br>Director as to which eye is operated first. |
|---|---|
| 915 | 4.7 Treatment during the Treatment Failure Identification Phase |
| 916 | After the 26 Week primary outcome visit, subjects will transition to the Treatment Failure |
| 917 | Identification Phase. Ongoing treatment will continue following the guidelines for the first six |
| 918 | months (26 weeks) as long as treatment failure criteria are not met at which time treatment will |
| 919 | be at the discretion of the Site Investigator. Investigators are urged to employ treatments from |
| 920 | another arm of the study before other treatments under these circumstances. |

| 921 | Chapter 5: Study Visits and Procedures |
|---|---|
| 922 | 5.1 Randomized Trial |
| 923 | 5.1.1 Study Visits and Phone Contacts |
| 924<br>925 | During the randomized trial, follow-up visits for all three groups will occur at weeks 4, 8 16, and $26 (\pm 7 \text{ days})$ timed from the day of randomization. |
| 926<br>927 | Post-operative visits may also be performed by the surgeon according to the surgeon's usual routine. |
| 928 | Additional office visits may occur as needed. |
| 929 | Phone contacts will occur at 12 and 20 weeks (±7 days). |
| 930 | 5.1.2 Safety Visits |
| 931<br>932<br>933<br>934<br>935<br>936 | Safety visits will occur in addition to study visits, with the timing dependent on the treatment group. The medical therapy only group generally will have visits 7 days and 14 days ( $\pm$ 4 days) following randomization whereas the surgery groups generally will have visits 7 days and 14 days ( $\pm$ 4 days) following each surgical procedure. Visit schedules can be modified at investigator discretion based on the participant's course and the 14-day visit could be skipped if there is substantial improvement in papilledema after 7 days. Additional visits can be scheduled as indicated. Reoperations at any time also will have a similar safety visit schedule. |
| 938 | 5.1.3 Study Visit Procedures |
| 939<br>940 | The following procedures will be performed for all subjects at each study visit, unless otherwise specified: |
| 941 | Medical/IIH history update |
| 942 | Adverse Events |
| 943 | Concomitant Medications |
| 944 | <ul> <li>Vital signs, including weight; (waist circumference at 26 Week only)</li> </ul> |
| 945 | Clinical Laboratories |
| 946 | • Refraction |
| 947 | Visual Acuity |
| 948 | Ocular Examination |
| 949 | <ul> <li>Metabolic Panel (16 and 26 Week only)</li> </ul> |
| 950 | • CBC (16 and 26 Week only) |
| 951 | • Humphrey visual field testing with 24-2 full-threshold program using size V stimulus |
| 952 | at 26 Week, two visual field examinations |

| 953<br>954 | At other study visits, one visual field examination will be done, but the VFRC may request the visual field examination be repeated |
|---|---|
| 955 | • Fundus Photographs |
| 956 | OCT* (optic nerve head and macula) |
| 957 | Dispense/prescribe acetazolamide and, if needed, furosemide |
| 958 | Drug Compliance/Accountability |
| 959 | Dietary counseling |
| 960 | <ul> <li>QoL questionnaires (26 Week only) – at study site or online</li> </ul> |
| 961 | • HIT-6 questionnaire (26 Week only) – at study site or online |
| 962 | • Lumbar puncture for CSF opening pressure measurement (26 Week; voluntary) |
| 963 | *The 26 Week OCT must be done <i>before</i> the lumbar puncture. |
| 964 | 5.1.4 Phone Contact Procedures |
| 965 | The Site Coordinator will contact the subject by telephone to review adverse events. |
| 966 | Medical/IIH History update |
| 967 | • Adverse Events |
| 968 | Review of Concomitant Medications |
| 969 | Review of Drug Compliance |
| 970 | Additional phone contacts, texts, and emails may be performed as needed. |
| 971 | 5.1.5 Safety Visit Procedures |
| 972 | The following procedures will be performed for all subjects at each safety visit: |
| 973 | Adverse Events |
| 974 | Concomitant Medications |
| 975 | <ul> <li>Vital signs, including weight</li> </ul> |
| 976 | • Refraction |
| 977 | Visual Acuity |
| 978 | Ocular Examination |
| 979 | • Humphrey Visual Field testing with 24-2 full-threshold program using size V stimulus |
| 980 | • OCT (optic nerve head and macula) |
| 981 | • Fundus Photographs (only at week 2) |
| 982 | Drug Compliance/Accountability |

| 983 | 5.2 Treatment Failure Identification Phase |
|---|---|
| 984 | 5.2.1 Follow-up Visits |
| 985<br>986 | Follow-up visits will occur at weeks 52 (12 months), 104 (2 years), and 156 (3 years) +4 weeks as long as the study is ongoing. |
| 987 | 5.2.2 Study Visit Procedures |
| 988 | Procedures at these visits will include the following: |
| 989 | Medical/IIH history update (includes all new treatments and adjustments of dosages) |
| 990 | Adverse Events |
| 991 | Concomitant Medications |
| 992 | Vital signs, including weight |
| 993 | • Refraction |
| 994 | Visual Acuity |
| 995 | Ocular Examination |
| 996 | • Humphrey Visual Field testing with 24-2 full-threshold program using size V stimulus |
| 997 | • Fundus Photographs |
| 998 | OCT (optic nerve head and macula) |
| 999 | Drug Compliance |
| 000 | <ul> <li>QoL questionnaires – at study site or online</li> </ul> |
| 001 | • HIT-6 questionnaire – at study site or online |
| 002<br>003 | If subject wants to discontinue birth control after the 6-month RCT, this should be discussed with the Site Investigator. |
| 004 | 5.2.3 Phone Contact Procedures |
| 005<br>006<br>007<br>008<br>009 | A phone, text or email contact will occur at 39 weeks by site staff. Subsequent contacts (every 3 months, starting at month 15 through month 33) will be by Coordinating Center staff for a structured interview to determine if IIH symptoms have worsened. If the caller has concerns about the subject, the site investigator will be notified and will be responsible for contacting the subject. |
| 010 | 5.3 Unscheduled Visits |
| 011<br>012<br>013<br>014 | An unscheduled visit can be performed at any time at investigator discretion, including the circumstance where the subject reports that IIH symptoms have worsened or if any unexpected adverse events develop. Testing performed and management decisions will be dependent on the circumstances of the visit and the findings |

| 1015 | 5.4 Extra Assessments for Subjects Who Appear to be Worsening |
|---|---|
| 1016<br>1017<br>1018<br>1019<br>1020<br>1021 | If a subject appears to be worsening, the subject will receive a combination of frequent contact (phone, text, email) and unscheduled visits. The Site Investigator will determine at the end of each visit whether the subject appears to be worsening clinically [guidelines being: 1) subject report of progressive visual loss, 2) papilledema is worsening, 3) OCT measures are worsening, 4) ETDRS acuity worsens more than 4 letters, or 5) PMD worsens more than 2 dB]. If the Site Investigator is unsure how to proceed, he/she will review the case with the Study co-Director. |
| 1022 | 5.5 Early Termination |
| 1023<br>1024 | For subjects who are withdrawing or being withdrawn from the study, a final visit should be scheduled as soon as possible. |
| 1025 | Procedures to be performed during the visit are the same as those listed in section 5.1.3. |
| 1026 | 5.6 Surgical Malfunction |
| 1027<br>1028<br>1029<br>1030<br>1031 | VPS and ONSF malfunction will be evaluated at every visit if symptoms and findings suggest it. If the Site Investigator, based on all clinical findings, believes that there may be a surgical procedure malfunction/failure, he/she will request an SMRC review. Similarly, if the Photo Reading Center or Visual Field Reading Center identify lack of improvement or worsening, a SMRC review can be triggered. |
| 1032 | 5.6.1 Criteria for SMRC Review |
| 1033 | Any of the below can trigger an SMRC review: |
| 1034 | 1. Either visual criteria for treatment failure are met (see section 5.7.1) |
| 1035<br>1036 | 2. Papilledema: failure of papilledema to improve from baseline or worsening of papilledema following improvement |
| 1037<br>1038 | 3. Site investigator believes there is substantial worsening of the subject's condition even if none of the other criteria are met |
| 1039 | 5.6.2 Surgical Malfunction Review by SMRC |
| 1040<br>1041<br>1042<br>1043<br>1044<br>1045<br>1046<br>1047<br>1048 | When triggered, the SMRC will review all available clinically-related information and reading center results to determine whether there is a non-disease associated cause (mechanical cause) for the lack of improvement or worsening. The site surgeon and investigator will participate in the review process as needed. The SMRC may request that certain exams be repeated for further evaluation. The evaluation for VPS may include a radionuclide shunt study. The evaluation for ONSF may consider orbital MRI or echography. If the SMRC believes a surgical malfunction is likely, the subject's surgical procedure will be evaluated to check the viability of the procedure. If the SMRC decides there was a problem with the surgery or a surgical device malfunction, they will discuss the case with the site investigator, the surgeon, and the Study co-Director (or committee member) to determine whether re-operation is indicated. |

| 1050<br>1051<br>1052 | The subject's safety is priority so if a site investigator or the SMRC Chair is confident a surgical malfunction occurred and emergent re-operation is needed, re-operation may be performed prior to full SMRC review. |
|---|---|
| 1053 | 5.6.3 Temporary Treatment Failure |
| 1054<br>1055<br>1056<br>1057<br>1058<br>1059<br>1060 | Temporary treatment failure is a situation that can occur in either of the surgical arms where the subject meets criteria for treatment failure (see section 5.7.1) and then has their surgical procedure revised or, in the case of ONSF, either revised or the other eye operated on. If the subject then recovers vision and no longer meets the criteria for treatment failure, they will continue the protocol treatment. If repeat surgery is not successful in improving vision out of the treatment failure criteria range, the case goes to the Adjudication Committee to determine if treatment failure has occurred. |
| 1061 | 5.7 Treatment Failure |
| 1062<br>1063<br>1064<br>1065<br>1066<br>1067<br>1068<br>1069 | Possible treatment failure will be evaluated at every visit if symptoms and findings suggest it. If the Site Investigator, based on all clinical findings, believes that there may be a treatment failure, the worsening will be confirmed with a repeat visual field examination (and ETDRS acuity testing if needed) on the same day or within four days of the original visual field. If the Visual Field Reading Center identifies lack of improvement or worsening, the site will be notified and repeat testing performed. If the worsening is confirmed (both visual field examinations having PMD that exceeds the cutoff value in 5.7.1 below), the case goes to the Adjudication Committee to determine if treatment failure has occurred. |
| 1070 | 5.7.1 Treatment Failure Criteria |
| 1071<br>1072 | If either of the below criteria for worsening are met, the subject will be considered for treatment failure by the Adjudication Committee: |
| 1073 | 1. Worsening of Full Threshold Size V 24-2 Perimetry. |
| 1074<br>1075 | a. Average baseline MD is equal to or better than -4 dB and visual function worsens more than 2 dB MD from the baseline average. |
| 1076<br>1077 | b. Average baseline MD is worse than -4 dB and equal to or better than -6 dB and visual function worsens more than 3 dB MD from baseline average. |
| 1078<br>1079 | <ul> <li>Average baseline MD is worse than -6 dB and visual function worsens more than 4 dB MD from baseline average.</li> </ul> |
| 1080 | 2. Worsening of 2 or more lines of ETDRS visual acuity |
| 1081 | 5.7.2 Treatment Failure Review by Adjudication Committee |
| 1082<br>1083<br>1084<br>1085<br>1086 | The Adjudication Committee will review possible treatment failures and determine if a treatment failure has occurred. The committee will be masked to treatment assignment and using all available clinically-related information, including fundus photo results, will decide whether the failure is most likely due to increased intracranial pressure or from another cause, such as perimetric artifact, poor subject effort, or the presence of another unrelated cause of visual loss. |

| 1087 | If the Adjudication Committee determines that a possible treatment failure is most likely due to |
|---|---|
| 1088 | IIH, the subject will be classified as having experienced a treatment failure. All cases that are |
| 1089 | sent to the Adjudication Committee will be reviewed first by the Study Director. If it is obvious |
| 1090 | that the patient meets criteria for treatment failure, they will be so designated. The case will |
| 1091 | subsequently be reviewed by the Adjudication Committee. |
| 1092 | When a subject meets the criteria for treatment failure, it is preferred that subsequent therapy |
| 1093 | come from one of the other two treatment arms but this decision will be deferred to the judgment |
| 1094 | of the Site Investigator. These subjects will continue to be followed at their set times for the full |
| 1095 | follow-up period (up to 3 years). The date of a confirmed treatment failure will be the date of the |
| 1096 | first visual field that triggered the Adjudication Committee review. |
| 1097 | If treatment failure is not confirmed, the subject will continue to follow his/her treatment group's |
| 1098 | protocol. |
| 1099 | |

# Figure 3. Algorithm for Review by Surgical Malfunction Review Committee

Criteria for Surgical Malfunction (Temporary TF):

- 1) Papilledema: at week 2 or after failure to improve from baseline or worsening following improvement
- 2) MD or ETDRS acuity worsening to TF levels
- 3) Site investigator worried there is a surgical malfunction

# SMRC reviews perimetry, OCT, disc photos, and clinical profile



1101

1102

1103

1104

1105

1106

1107

1108 1109

1110

#### 5.7.3 Visit Schedule Once Treatment Failure is Reached

When a subject reaches treatment failure prior to the 6 Month visit window, the subject should be brought back as soon as possible for an unscheduled visit and all 6 Month visit procedures should be performed. The subject should be directed to remain on medical therapy (if on medical therapy) until seen for this visit, unless instructed otherwise by the Site Investigator. The subject should then return for the scheduled 6 Month visit and then the 12 Month visit. After the 12 Month visit, subjects will then continue in the Treatment Failure Identification Phase of the study with annual visits.

| 1111<br>1112 | Chapter 6: Testing Procedures, Questionnaires, Clinical Assessments, and Laboratory Testing |
|---|---|
| 1113 | 6.1 Testing Procedures |
| 1114 | The testing procedures are noted below and details are provided in the Site Procedures Manual. |
| 1115 | 6.2 Intraocular Pressure |
| 1116 | Intraocular pressure will be measured using Goldmann tonometry. |
| 1117 | 6.3 Refraction and Visual Acuity |
| 1118<br>1119<br>1120 | At each protocol visit, a standardized refraction will be performed in both eyes. This will be followed by testing of visual acuity using ETDRS charts. Both will be administered by a certified technician masked to treatment group as best as possible. |
| 1121<br>1122<br>1123 | Although it is not possible to fully mask the technician to whether or not a subject had ONSF, all subjects will wear hairnest during the testing after randomization through the Week 8 visit in order to provide masking to VPS. |
| 1124 | 6.4 Papilledema Grading |
| 1125 | Site investigators will be trained to grade papilledema using the Frisén scale. <sup>77</sup> |
| 1126<br>1127<br>1128 | Fundus photography: Digital fundus photographs centered on the optic disc will be taken at each visit. The severity of papilledema will be graded by the Photography Reading Center (PRC) using the Frisén scale. <sup>77,78</sup> |
| 1129 | 6.5 Perimetry |
| 1130<br>1131<br>1132 | Automated perimetry will be performed using the Humphrey Field Analyzer (HFA) 24-2 full-threshold program using a size V stimulus in both eyes by a certified technician masked as best as possible to treatment group. The MOP provides a detailed description of this procedure. |
| 1133<br>1134<br>1135<br>1136<br>1137 | Although it is not possible to fully mask the visual field technician to whether or not a subject had ONSF, all subjects will wear hairnest during the visual field examination after randomization through the Week 8 visit in order to provide masking to VPS. The use of a standardized visual field protocol should limit the influence of the visual field technician on the results of the examination. |
| 1138 | 6.6 OCT |
| 1139<br>1140<br>1141<br>1142 | Spectral-domain OCT evaluations of the optic nerves, peripapillary RNFL, and macula will be obtained using a Cirrus <sup>™</sup> (Carl Zeiss-Meditec, Inc, Dublin, CA) or Spectralis <sup>®</sup> (Heidelberg Engineering, Inc, Carlsbad, CA) spectral-domain OCT. The subject must have the same brand of OCT machine used for data collection at each visit. |

| 1143 | 6.7 Lumbar Puncture |
|---|---|
| 1144<br>1145<br>1146 | Lumbar puncture is performed as part of usual care at baseline. Although repeat lumbar puncture is not considered standard of care, subjects will undergo a second voluntary lumbar puncture for CSF opening pressure measurement at the 6-month visit, following the procedure detailed in the |
| 1147 | MOP. |
| 1148 | 6.8 Quality of Life Assessment |
| 1149<br>1150 | The NEI VFQ-25 and the 10-item Neuro-ophthalmic Supplement to the VFQ-25 will be used, as well as the SF-36v2. <sup>79</sup> Testing time is approximately 20 minutes. |
| 1151 | 6.9 Headache Disability Rating |
| 1152<br>1153<br>1154 | Headache disability will be rated using the HIT-6 (Headache Impact Test), <sup>80</sup> a 6-item scale that is commonly used to rate migraine disability and has been validated for IIH. Testing time is 1-2 minutes. |
| 1155 | 6.10 Neurologic and Physical Examination |
| 1156<br>1157 | A standard neurological evaluation will be performed at screening. When indicated, a general medical examination will be performed. |
| 1158 | 6.11 Clinical Laboratory Tests |
| 1159 | CBC with platelet count will be obtained at Baseline and at Weeks 16 and 26 for all subjects. |
| 1160<br>1161 | A comprehensive metabolic profile, including liver function tests, electrolytes, and amylase, will be obtained at Baseline and at Weeks 16 and 26 for all subjects. |
| 1162 | For subjects taking furosemide, serum potassium and sodium levels will be checked prior to each |
| 1163 | dosage change, after reaching the maximum tolerated dosage, and then at each subsequent visit. |
| 1164 | This testing will be performed at a local laboratory. |
| 1165 | Routine clinical laboratory tests will be performed locally by the site or the subject's local |
| 1166 | laboratory if travel to the site is not convenient. The Site Investigator will review the laboratory |
| 1167 | values. The Site Investigator will prescribe appropriate supplementation for hypokalemia, |
| 1168 | hyponatremia and symptomatic bicarbonate deficiency, and may enlist the help of the subject's |
| 1169 | primary physician to help manage abnormal laboratory results, if necessary. |

| 1170 | Chapter 7: Adverse Event Reporting |
|---|---|
| 1171 | 7.1 Adverse Events |
| 1172 | 7.1.1 Definitions |
| 1173<br>1174<br>1175 | Adverse Event (AE): Any untoward medical occurrence in a study subject, irrespective of the relationship between the adverse event and the study drug or surgery (see 7.1.2 for what adverse events require reporting in this protocol). |
| 1176 | Serious Adverse Event (SAE): Any untoward medical occurrence that: |
| 1177 | • Results in death. |
| 1178<br>1179 | • Is life-threatening; (a non-life-threatening event which, had it been more severe, might have become life-threatening, is not necessarily considered a serious adverse event). |
| 1180 | <ul> <li>Requires inpatient hospitalization or prolongation of existing hospitalization.</li> </ul> |
| 1181<br>1182 | <ul> <li>Results in persistent or significant disability/incapacity or substantial disruption of the<br/>ability to conduct normal life functions.</li> </ul> |
| 1183 | • Is a congenital anomaly or birth defect. |
| 1184<br>1185<br>1186 | • Is considered a significant medical event by the investigator based on medical judgment (e.g., may jeopardize the subject or may require medical/surgical intervention to prevent one of the outcomes listed above). |
| 1187 | 7.1.2 Reporting Adverse Events |
| 1188<br>1189<br>1190 | Symptoms and signs, including visual symptoms and headaches, that are considered to be due to IIH will be captured on a visit/phone case report form and are not considered to be adverse events unless SAE criteria are met. |
| 1191<br>1192<br>1193<br>1194<br>1195<br>1196 | Certain adverse events that are known side effects of acetazolamide and furosemide will be captured on a visit/phone case report form (including paresthesia, dizziness, nausea, vomiting, diarrhea, loss of appetite, acid reflux, skin rash, dyspnea, hypercapnia, depression, anxiety, tinnitus, fatigue) for all subjects, regardless of whether taking study medication. A separate Adverse Event Form is only completed for these specific events if SAE criteria are met or the event was severe enough that it resulted in discontinuation of study drug. |
| 1197<br>1198<br>1199 | Expected symptoms post-surgery will be captured on a visit/phone case report form. A separate Adverse Event Form is only completed for these specific events if SAE criteria are met or if the onset date is outside the expected duration of occurrence post-surgery, regardless of intensity. |
| 1200<br>1201<br>1202 | Laboratory results of interest will be recorded on a laboratory data case report form. A separate Adverse Event Form is only completed for laboratory abnormalities that are considered clinically significant by the investigator. |

| 1203<br>1204<br>1205 | During the first 6 months, all other events (not described above) meeting the definition of adverse event will be reported on an Adverse Event Form. After the first 6 months, only those events meeting SAE criteria will be reported on an Adverse Event Form. |
|---|---|
| 1206 | 7.1.3 Relationship of Adverse Event to Study |
| 1207<br>1208<br>1209<br>1210 | The study investigator will assess the relationship of any adverse event reported on an Adverse Event Form to be related or unrelated to a study intervention or procedure by determining if there is a reasonable possibility that the adverse event may have been caused by the intervention or procedure. |
| 1211<br>1212 | To ensure consistency of adverse event causality assessments, investigators should apply the following general guideline when determining whether an adverse event is related: |
| 1213 | <u>Yes</u> |
| 1214<br>1215<br>1216<br>1217<br>1218<br>1219 | There is a plausible temporal relationship between the onset of the adverse event and the study intervention/procedure, and the adverse event cannot be readily explained by the subject's clinical state, intercurrent illness, or concomitant therapies; and/or the adverse event follows a known pattern of response to the study intervention/procedure; and/or the adverse event abates or resolves upon discontinuation of the study intervention/procedure or dose reduction and, if applicable, reappears upon re-challenge. |
| 1220 | <u>No</u> |
| 1221<br>1222<br>1223<br>1224 | Evidence exists that the adverse event has an etiology other than the study intervention/procedure (e.g., preexisting medical condition, underlying disease, intercurrent illness, or concomitant medication); and/or the adverse event has no plausible temporal relationship to study intervention/procedure. |
| 1225 | 7.1.4 Intensity of Adverse Events |
| 1226<br>1227<br>1228<br>1229 | The intensity of an adverse event will be rated on a three-point scale: (1) mild, (2) moderate, or (3) severe. It is emphasized that the term severe is a measure of intensity; thus, a severe adverse event is not necessarily serious. For example, itching for several days may be rated as severe, but may not be clinically serious. |
| 1230<br>1231 | • MILD: Usually transient, requires no special treatment, and does not interfere with the subject's daily activities. |
| 1232<br>1233<br>1234 | <ul> <li>MODERATE: Usually causes a low level of inconvenience or concern to the subject and<br/>may interfere with daily activities, but is usually ameliorated by simple therapeutic<br/>measures.</li> </ul> |
| 1235<br>1236 | • SEVERE: Interrupts a subject's usual daily activities and generally requires systemic drug therapy or other treatment. |
| 1237 | 7.1.5 Coding of Adverse Events |
| 1238 | Adverse events will be coded using the MedDRA dictionary |

| 1239 | 7.1.6 Outcome of Adverse Event |
|---|---|
| 1240 | The outcome of each reportable adverse event will be classified by the investigator as follows: |
| 1241<br>1242 | • RECOVERED/RESOLVED: The subject recovered from the AE/SAE without sequelae. Record the AE/SAE stop date. |
| 1243<br>1244 | • RECOVERED/RESOLVED WITH SEQUELAE: The event persisted and had stabilized without change in the event anticipated. Record the AE/SAE stop date. |
| 1245<br>1246 | <ul> <li>NOT RECOVERED/NOT RESOLVED: An ongoing AE/SAE is defined as the event<br/>was ongoing with an undetermined outcome.</li> </ul> |
| 1247<br>1248 | <ul> <li>An ongoing outcome will require follow-up by the site in order to determine the final<br/>outcome of the AE/SAE.</li> </ul> |
| 1249<br>1250<br>1251 | <ul> <li>The outcome of an ongoing event at the time of death that was not the cause of death,<br/>will be updated and recorded as "resolved" with the date of death recorded as the stop<br/>date.</li> </ul> |
| 1252<br>1253<br>1254<br>1255 | • FATAL: A fatal outcome is defined as the SAE that resulted in death. Only the event that was the cause of death should be reported as fatal. AEs/SAEs that were ongoing at the time of death; however, were not the cause of death, will be recorded as "resolved" at the time of death. |
| 1256<br>1257<br>1258 | • UNKNOWN: An unknown outcome is defined as an inability to access the subject or the subject's records to determine the outcome (for example, a subject that was lost to follow-up). |
| 1259<br>1260<br>1261<br>1262<br>1263 | All clinically significant abnormalities of clinical laboratory measurements or adverse events occurring during the study and continuing at study termination should be followed by the subject's physician and evaluated with additional tests (if necessary) until diagnosis of the underlying cause, or resolution. Follow-up information should be recorded on source documents. |
| 1264<br>1265<br>1266<br>1267<br>1268 | If any reported adverse events are present when a subject completes the study, or if a subject is withdrawn from the study due to an adverse event, the subject will be contacted for re-evaluation within 2 weeks. If the adverse event has not resolved, additional follow-up will be performed as appropriate. Every effort should be made by the Investigator or delegate to contact the subject until the adverse event has resolved or stabilized. |
| 1269 | 7.2 Pregnancy Reporting |
| 1270<br>1271 | If pregnancy occurs during the 6-month RCT, study drug will be discontinued. The occurrence of pregnancy will be reported on an AE Form. |
| 1272 | 7.3 Timing of Event Reporting |
| 1273<br>1274 | Serious, unexpected treatment-related adverse events must be reported to the Coordinating Center within 24 hours via completion of the online serious adverse event form. |
| 1275<br>1276 | Other reportable adverse events as defined in section 7.1.2 will be reported within 3 days of the investigator becoming aware of the event by completion of an electronic case report form. |

| 1277<br>1278<br>1279 | The Coordinating Center will notify all participating investigators of any adverse event that is serious, related, and unexpected. Notification will be made within 10 working days after the Coordinating Center becomes aware of the event. |
|---|---|
| 1280<br>1281<br>1282 | Each principal investigator is responsible for reporting serious study-related adverse events and abiding by any other reporting requirements specific to his/her Institutional Review Board or Ethics Committee. |
| 1283 | The sponsor will report any serious, unexpected treatment-related adverse events to the FDA. |
| 1284 | |
| 1285 | 7.4 Stopping Criteria |
| 1286 | 7.4.1 Subject Discontinuation of Study Drug |
| 1287 | Rules for discontinuing study drug use are described below. |
| 1288<br>1289<br>1290<br>1291 | • The investigator believes it is unsafe for the subject to continue to receive the drug. This could be due to the development of a potential side effect of the drug, a new medical condition or worsening of an existing condition; or subject behavior contrary to the indications for use of the drug that imposes on the subject's safety |
| 1292 | <ul> <li>The subject requests that the treatment be stopped</li> </ul> |
| 1293<br>1294 | • Subject pregnancy during 6-month RCT (discontinuation at investigator discretion during Treatment Failure Identification Phase) |
| 1295<br>1296 | Even if the study drug is discontinued, the subject will be encouraged to remain in the study through the final study visit. |
| 1297 | 7.5 Medical Monitor |
| 1298<br>1299 | A Medical Monitor will review all reported adverse events reported on an Adverse Event Form, solicited events captured on a visit/phone case report form, and laboratory abnormalities. |
| 1300<br>1301<br>1302 | The Medical Monitor will assess each event for appropriate coding of intensity, criteria for SAE, relationship to study drug/procedure, and MedDRA classification. The Medical Monitor's coding will be considered final. |
| 1303 | 7.6 Independent Safety Oversight |
| 1304<br>1305<br>1306<br>1307 | A Data and Safety Monitoring Committee (DSMC), selected by the National Eye Institute, will provide study oversight. The Committee will be sent serious, unexpected, treatment-related adverse events for expedited review and all adverse events in a cumulative report approximately every 6 months. |
| 1308 | 7.7 Criteria for Suspending or Terminating Overall Study |
| 1309<br>1310 | There are no pre-specified criteria for suspending or terminating the study. Such decisions will be made by the DSMC based on their review of accumulated safety data. |

| 1311 | Chapter 8: Miscellaneous Considerations |
|---|---|
| 1312 | 8.1 Subject Compensation |
| 1313 | Subject compensation will be specified in the informed consent form. |
| 1314 | 8.2 Subject Withdrawal |
| 1315<br>1316<br>1317 | Participation in the study is voluntary, and a subject may withdraw at any time. For subjects who withdraw, their data will be used up until the time of withdrawal. If possible, a final visit will be completed for all subjects who are terminating the study early (see section 5.5). |
| 1318<br>1319 | A subject may be withdrawn from the study at the discretion of the Site Investigator or the Study co-Director for the following reasons: |
| 1320 | • Adverse event, but only if follow-up presents a risk to the subject's safety |
| 1321<br>1322 | <ul> <li>Noncompliance with study medications, but only if follow-up presents a risk to the<br/>subject's safety</li> </ul> |
| 1323 | • Development of a condition, but only if follow-up presents a risk to the subject's safety |
| 1324<br>1325 | Prior to withdrawing subject from the study, the Site Investigator must contact the Study co-<br>Director to discuss the case. |
| 1326 | 8.3 Confidentiality |
| 1327<br>1328<br>1329<br>1330<br>1331 | For security and confidentiality purposes, subjects will be assigned an identifier that will be used instead of their name. Protected health information gathered for this study will be shared with the coordinating center, the Jaeb Center for Health Research in Tampa, FL and the enrollment center, Mount Sinai in New York, NY. De-identified subject information may also be provided to research sites involved in the study. |

| 1332 | <b>Chapter 9: Statistical Consideration</b> |
|---|---|
| 1333 | 9.1 Statistical and Analytical Plans |
| 1334<br>1335<br>1336 | The approach to sample size and statistical analyses are summarized below. A detailed statistical analysis plan will be written and finalized prior to viewing any outcome data. The analysis plan synopsis in this chapter contains the framework of the anticipated final analysis plan. |
| 1337 | 9.2 Intention-to-Treat Principle |
| 1338<br>1339<br>1340<br>1341<br>1342<br>1343<br>1344<br>1345 | The primary statistical analyses for this trial will be performed according to the intention-to-treat principle and will include all randomized subjects and eligible eyes. Every effort will be made to retain subjects in this study, to promote adherence to the study protocol, and to collect all data at every visit. If a subject cannot tolerate study medication or refuses to receive the study intervention, we will continue to follow and evaluate that subject if he/she is willing. If a subject drops out, attempts will be made to bring the subject back for a final evaluation. Compliance with trial procedures, drop-outs/drop-ins, and reasons for subject withdrawal will be carefully tracked throughout the study. |
| 1346 | 9.3 Analysis of the Primary Outcome Variable |
| 1347 | 9.3.1 Primary Statistical Model |
| 1348<br>1349<br>1350<br>1351<br>1352<br>1353<br>1354<br>1355 | The primary outcome variable will be the change from baseline to the first of Month 6 or time of treatment failure in PMD in an eligible eye, with data from all eligible eyes included in the primary analysis. The primary statistical analysis will involve fitting an analysis of covariance model using generalized estimating equations (GEE) with treatment group as the factor of interest and baseline PMD as a covariate. These analyses will accommodate correlation among the within-subject responses between the two eyes; an exchangeable working correlation structure will be used. Standard errors for the model parameters will be estimated using the robust "sandwich" estimators. The model also does not rely on the assumption of normality. |
| 1356<br>1357<br>1358<br>1359<br>1360<br>1361<br>1362 | This model will be used to determine Bonferroni-adjusted confidence intervals for the three pairwise differences among the adjusted treatment group mean responses (treatment effects); likewise, tests will be performed to compare the adjusted treatment group means using a Bonferroni-adjusted two-tailed significance level. An overall confidence coefficient of 98.3% and corresponding significance level of 1.7% for each comparison will be maintained, but as discussed in section 9.8.2 below, the confidence coefficient for interval estimation and significance level for hypothesis testing will be adjusted for the interim analysis for efficacy. |
| 1363<br>1364<br>1365<br>1366<br>1367<br>1368<br>1369<br>1370 | Treatment of subjects who have reached criteria for treatment failure will be at the discretion of the Site Investigator, and this treatment may yield a different outcome than randomized treatment (investigators are urged to employ treatments from another arm of the study before other treatments under these circumstances). For this reason, the primary outcome variable for subjects who reach criteria for treatment failure prior to Month 6 will be the PMD measured at the time of treatment failure for purposes of the primary analysis. It is anticipated that no more than 15% of subjects will reach criteria for treatment failure prior to Month 6. As the most important of the secondary outcome variable analyses, A secondary outcome analysis will be performed that will |

1371 include the PMD for these subjects that was obtained at Month 6, regardless of treatment received after treatment failure. 1372 1373 9.3.2 Adjustment for Baseline Characteristics 1374 If clinically important differences are found between the groups at baseline, particularly with 1375 regard to important variables such as age, gender, race/ethnicity, or visual acuity, the primary 1376 outcome analyses will be repeated after statistically adjusting for these differences. These 1377 analyses will be considered secondary, however. 1378 9.3.3 Investigation of Treatment by Covariate Interactions 1379 We will investigate the interaction between treatment group and selected baseline covariates 1380 (age, race/ethnicity, PMD, papilledema grade, RNFL thickness, total retinal thickness, optic nerve head volume, visual acuity, presence of transient visual obscurations, and the symptom of 1381 1382 constant visual loss) separately by adding the appropriate main effect and interaction terms to the 1383 primary statistical model and testing for significance of the interaction. Since the power to detect potentially meaningful interactions will be limited, the magnitudes of mean responses to 1384 1385 treatment in the relevant subgroups will be examined. The observation of clinically important 1386 subgroup differences in mean treatment response will serve as hypothesis generation for possible 1387 future studies designed to address specifically the issue of differential therapeutic response. 1388 Although these analyses are purely exploratory, those involving papilledema grade, PMD, visual 1389 acuity, and race/ethnicity will be given higher priority. 1390

### 9.3.4 Verification of Model Assumptions

The underlying assumptions of the statistical model to be used in the primary analysis will be thoroughly checked (e.g., linearity), and remedial measures (e.g., transformations) may be taken if serious violations of these assumptions are detected.

#### 9.3.5 Treatment of Missing Data

1391

1392

1393

1394

1395

1396

1397

1398

1399

1400

1401

1402

1403

1404

1405

1406

1407

1408

1409 1410

1411

1412

Multiple imputation will be used to deal with missing data. This will be applied using a regression-based imputation model. For subjects with complete data up to a particular visit, a multiple regression model will be fit that includes the outcome at that visit as the dependent variable and outcomes at previous visits and treatment group as independent variables. Separate models will be similarly constructed for each visit (Weeks 1, 4, 8, 16, and 26). Using these regression models, a missing value for a subject at a particular visit will be imputed as a draw from the predictive distribution given the outcomes at previous visits (some possibly imputed) and treatment group. This will be done sequentially starting with the Week 1 visit and ending with the Week 26 (Month 6) visit. This process will be repeated 100 times, resulting in 100 complete analysis data sets. The analyses will be performed separately for each of the 100 complete analysis data sets, and the results will be combined into one multiple imputation inference (estimated treatment effect and associated confidence interval and p-value) using Rubin's rules. 93,94 This approach is appropriate for data sets that have a monotone missing data pattern. If the data set does not precisely have this pattern, the monotone data augmentation method using Markov-Chain Monte-Carlo 95,96 will be used to impute the small amount of missing data that is required to make the missing data pattern monotone before applying the multiple imputation algorithm described above. This approach should accommodate missing data in an appropriate way under the missing at random (MAR) assumption. 88,89

| 1413<br>1414<br>1415<br>1416<br>1417<br>1418<br>1419<br>1420<br>1421<br>1422 | Separate secondary analyses may also be performed that, for example, may group subjects according to treatment actually received (whether or not this was the randomly assigned treatment) and/or exclude subjects who had incomplete follow-up, took less than a certain threshold of their medication, or had another major protocol violation. The identification of subjects to be excluded from these analyses will be determined before the masking is broken (i.e., before data analysis). Of course, such analyses may lead to biased estimates of the actual treatment effects, but they may provide an indication of the sensitivity of the analyses to drop-ins/drop-outs and noncompliance. Methods such as those based on propensity score stratification or inverse probability weighting can be employed in this setting in which non-randomized groups are to be compared. |
|---|---|
| 1423 | 9.4 Analysis of the Secondary Outcome Variables for Efficacy |
| 1424<br>1425<br>1426<br>1427<br>1428 | The most important secondary outcome variable for efficacy will be change from baseline to Month 6 in PMD in an eligible eye, with data from all eligible eyes included in this analysis. This is in contrast to the primary outcome variable for efficacy that is change in PMD from baseline to the first of Month 6 or time of treatment failure in an eligible eye, with data from all eligible eyes included in this analysis. |
| 1429<br>1430<br>1431<br>1432<br>1433<br>1434<br>1435<br>1436<br>1437 | The following additional secondary outcome variables will be evaluated at six months: change in CSF opening pressure measurement by lumbar puncture; change in papilledema grade (PRC and Site Investigator); changes in OCT measures (RNFL thickness, total retinal thickness, optic nerve head volume, ganglion cell layer thickness, optic nerve canal shape); changes in ETDRS visual acuity scores; changes in QoL assessments (SF-36, VFQ-25 and its 10-item supplement), changes in headache assessments (HIT-6 Inventory and headache severity); Visual Field Reading Center (VFRC) determination by three visual field experts of whether the visual field examination has improved, remained the same, or worsened; treatment failure; and surgical failure (transient or otherwise depending on attempts to repair malfunctions). |
| 1438<br>1439<br>1440<br>1441 | With the exception of CSF opening pressure, these outcome variables will also be examined at Months 12, 24, and 36. Of special interest is the outcome of time from randomization to treatment failure. Time from randomization to failure due to surgical malfunction (even if temporary) is also of interest in the long-term follow-up phase. |
| 1442<br>1443<br>1444<br>1445<br>1446<br>1447 | Treatment effects on secondary outcome variables for efficacy that are continuous will be analyzed using the same methods described above for the primary outcome variable, except that a working correlation structure will not be needed for variables that are not eye-specific. Variables to be analyzed in this manner include CSF opening pressure, OCT measures, quality of life as measured by the NEI-VFQ-25 + 10-item neuro-ophthalmic supplement and the SF-36, headache disability (HIT-6 Inventory), and headache severity. |
| 1448<br>1449<br>1450<br>1451 | The model will be used to determine Bonferroni-adjusted 98.3% confidence intervals for the three pair-wise differences among the adjusted treatment group mean responses (treatment effects) at Month 6; likewise, tests will be performed to compare the adjusted treatment group means at Month 6 using a Bonferroni-adjusted two-tailed significance level of 1.7%. |
| 1452<br>1453 | For categorical outcome variables that are dichotomous (e.g., presence of headache, surgical failure) or ordinal (visual field examination ratings by the VFRC, graded as improved, no |

| 1454<br>1455 | change, or worse), logistic regression models (or proportional odds models for ordinal outcomes) will be used to assess treatment effects. These models will include treatment group as the factor |
|---|---|
| 1456 | of interest and the baseline value of the outcome variable (for presence of headache) or baseline |
| 1457 | PMD (for surgical failure) as covariates. Likelihood-ratio tests will be performed for significance |
| 1458 | of the adjusted treatment group odds ratios representing pair-wise treatment group comparisons, |
| 1459 | and 98.3% confidence intervals will be constructed for these odds ratios. Other aspects of the |
| 1460<br>1461 | analysis of the primary outcome variable (e.g., further adjustment for baseline factors, |
| 1401 | examination of interactions, verification of model assumptions) will also be considered. |
| 1462 | For dichotomous outcomes that are measured repeatedly over time (e.g., presence of headache), |
| 1463 | if a subject is missing a response at a particular visit, missing data will be imputed using logistic |
| 1464 | regression-based multiple imputation. <sup>93</sup> For subjects with complete data up to a particular visit, a |
| 1465 | logistic regression model will be fit that includes the outcome at that visit as the dependent |
| 1466 | variable and outcomes at previous visits and treatment group as independent variables. Separate |
| 1467 | models will be similarly constructed for each visit. Using these logistic regression models, a |
| 1468 | missing value for a subject at a particular visit will be imputed as a draw from the predictive |
| 1469 | distribution given the outcomes at previous visits (some possibly imputed) and treatment group |
| 1470 | of the subject. This will be done sequentially starting with the Week 1 visit and ending with the |
| 1471 | Month 6 visit. This process will be repeated 100 times, resulting in 100 complete analysis data |
| 1472<br>1473 | sets. The analyses will be performed separately for each of the 100 complete analysis data sets, |
| 1473 | and the results will be combined into one multiple imputation inference (estimated odds ratios [treatment effects] and associated confidence intervals and p-values) using Rubin's rules. 93,94 |
| 14/4 | [treatment effects] and associated confidence intervals and p-values) using Rubin's futes. |
| 1475 | 9.5 Compliance Outcomes |
| 1476 | Data concerning compliance with acetazolamide (pill counts, serum bicarbonate levels) and |
| 1477 | surgical therapy will be summarized by treatment group and visit. Subjects with two eligible |
| 1478 | eyes will have this information summarized by eye as well as by treatment group and visit. |
| 1479 | Change in weight will be used as a summary of compliance with diet. |
| 1480 | 9.6 Analysis of Safety and Tolerability Outcomes |
| 1481 | 9.6.1 Adverse Events |
| 1482 | All reportable adverse events will be tabulated by treatment group in a listing of each reported |
| 1483 | Medical Dictionary for Regulatory Activities (MedDRA) term and summarized over each |
| 1484 | MedDRA System Organ Class. Details will be provided in a listing of each event. |
| 1485<br>1486 | In addition, the following will be tabulated by treatment group. When applicable, events will be tabulated by eye within person: |
| 1700 | tabulated by eye within person. |
| 1487 | <ul> <li>Number of adverse events</li> </ul> |
| 1488 | <ul> <li>Number of subjects with at least one event</li> </ul> |
| 1489 | <ul> <li>Number of serious adverse events</li> </ul> |
| 1490 | <ul> <li>Number of subjects with at least one serious adverse event</li> </ul> |
| 1491 | <ul> <li>Number of hospitalizations and reasons for the hospitalization</li> </ul> |

| 1492 | <ul> <li>Number of adverse events thought by investigator to be related to study drug</li> </ul> |
|---|---|
| 1493 | • Number of subjects who stopped the intervention in response to an adverse event |
| 1494<br>1495 | For binary variables, Fisher exact tests will be used to compare treatment groups. For counts, groups will be compared using Poisson regression. |
| 1496<br>1497<br>1498<br>1499<br>1500<br>1501 | For each adverse event, the treatment groups will be compared in a pair-wise fashion regarding the occurrence of at least one event using Fisher's exact tests; numbers of individual events will also be described. The comparisons will be repeated excluding all mild symptoms. Similar analyses will be performed after grouping adverse events by body system using Medical Dictionary for Regulatory Activities (MedDRA) coding. All subjects will be included in these analyses. |
| 1502 | 9.6.2 Tolerability Outcomes |
| 1503<br>1504<br>1505<br>1506<br>1507 | Tolerability will be primarily measured by ability to complete 6 months of follow-up on the originally assigned treatment. A complete accounting of subject disposition will be summarized by treatment group, including a tabulation of subject withdrawals, dosage reductions/ discontinuations of study medication due to adverse events (with reasons for each), receipt of surgery other than that randomly assigned, and surgical failures. |
| 1508 | 9.6.3 Laboratory Test Results and Vital Signs |
| 1509<br>1510<br>1511 | Continuous measures of safety such as laboratory test results (e.g., CBC with platelet count, electrolytes, potassium, bicarbonate, and liver function tests) and vital signs and anthropometric measures (e.g., blood pressure, weight, and waist circumference) will be analyzed descriptively. |
| 1512<br>1513 | Proportions of subjects with particular laboratory test abnormalities will be compared between the treatment groups in a pair-wise fashion using Fisher's exact tests. |
| 1514 | 9.7 Analysis of Long-Term Follow-Up Data |
| 1515<br>1516<br>1517<br>1518<br>1519<br>1520<br>1521<br>1522<br>1523<br>1524<br>1525<br>1526 | An important set of analyses will consider the outcome of time from randomization to treatment failure. The statistical analysis of this outcome variable will involve fitting a Cox proportional hazards regression model with treatment group as the factor of interest and baseline PMD in the best eligible eye as a covariate. This model will be used to determine Bonferroni-adjusted 98.3% confidence intervals for the adjusted hazard ratios for the three pair-wise treatment group comparisons; likewise, likelihood ratio tests will be performed for significance of these hazard ratios using a Bonferroni-adjusted two-tailed significance level of 1.7%. Kaplan-Meier curves will be used to describe the cumulative probability of treatment failure over time in each treatment group. For subjects who do not experience treatment failure, event times will be censored at the last subject contact at which the subject was determined to not have experienced treatment failure (e.g., at the time of premature withdrawal from the trial or at the final trial visit). |
| 1527<br>1528<br>1529 | As described above for the primary outcome variable for efficacy, secondary analyses of time to treatment failure that adjust for additional baseline covariates may be considered depending on the comparability of the treatment groups at baseline, and examination of interactions between |

| 1530<br>1531 | treatment group and selected baseline covariates will be performed using the Cox proportional hazards model. |
|---|---|
| 1532<br>1533<br>1534<br>1535<br>1536<br>1537<br>1538<br>1539<br>1540<br>1541<br>1542 | The underlying assumptions of the Cox proportional hazards models will be checked and a thorough analysis of the martingale residuals and other diagnostics will be performed $^{102}$ . Remedial measures (e.g., covariate transformation) will be taken if serious violations of these assumptions are detected. The proportional hazards assumption will be assessed graphically by plotting $\log(-\log(\hat{S}(t)))$ vs. $\log(time)$ for each of the treatment groups, and by plots of smoothed Schoenfeld residuals $^{101}$ . This assumption will also be examined by dividing the time scale into 6-month periods and estimating the treatment group hazard ratios separately in each of these periods through the use of time-dependent covariates $^{103}$ . The period length of 6 months may be adjusted prior to unmasking, based on the observed distribution of event times, if relatively few events occur during 6-month periods. Treatment group comparisons will be described in this manner if the proportional hazards assumption appears to be seriously violated. |
| 1543<br>1544<br>1545<br>1546<br>1547 | An additional important assumption of the methods to be used to analyze time to treatment failure is the independence between the censoring time and the (unobserved) event time. Sensitivity analyses will be performed that treat subjects with event times that are censored prior to their scheduled end of follow-up as having experienced the event a short time (one week) after censoring. |
| 1548<br>1549<br>1550<br>1551<br>1552<br>1553<br>1554<br>1555 | Analyses of the primary and secondary outcome variables for efficacy using data collected after the 6-month visit will be analyzed according to the initial treatment strategy using the same methods described above. This will include surgical procedure complications or transient malfunctions. More complex analyses may be performed that take into account the introduction of other treatments (e.g., surgery in those assigned to medical therapy) depending on how often this occurs. It will necessarily be difficult to make inferences about the effectiveness of subsequent treatments; however, analyses using marginal structural models 100,104 may prove useful for this purpose. Outcomes such as surgical failure and IIH recurrence (in those whose vision is initially restored) will be summarized descriptively over time. |
| 1557 | 9.8 Interim Analyses |
| 1558 | 9.8.1 Interim Analyses for Safety |
| 1559<br>1560<br>1561<br>1562<br>1563<br>1564<br>1565<br>1566<br>1567<br>1568<br>1569 | Interim analyses of safety data will be performed periodically throughout the trial. While the safety of subjects will be the primary concern of the DSMC, it is difficult to formulate precise stopping guidelines that would cover all of the possible situations that might arise. Adverse events, particularly serious adverse events and surgical complications, will have to be considered carefully by the DSMC in terms of treatment group imbalances and severity. Events of particular concern include the following: death, absence of light perception, hypokalemia (from Lasix use), surgery-associated visual loss (from either VPS or ONSF), fenestration failure and orbital infection (from ONSF), and shunt failure, infection, seizures, and subdural hematoma (from VPS). If potential safety concerns are identified, the DSMC may require review of visual field data in order to evaluate the risk-benefit of continuing the trial as planned or modifying (or halting) the trial. |

| 15/0 | 9.8.2 Interim Analyses for Efficacy |
|---|---|
| 1571<br>1572<br>1573<br>1574<br>1575<br>1576 | We propose to perform a single interim analysis for efficacy based on the primary outcome efficacy variable. This will be performed after 50% of the subjects have completed (or were scheduled to have completed, based on their randomization date) their Month 6 visit and will only include data from these 50% of subjects. Given that recruitment of the 180 subjects will take place over 3 years, assuming that recruitment is uniform over time, it is anticipated that slightly fewer than 70% of the subjects will be enrolled at the time of the interim analysis. |
| 1577<br>1578<br>1579<br>1580<br>1581<br>1582<br>1583<br>1584<br>1585<br>1586<br>1587<br>1588<br>1589 | The analysis will involve pair-wise comparisons among the treatment groups with respect to the primary outcome efficacy variable; the significance level used for each comparison will be that determined by an O'Brien-Fleming $\alpha$ -spending function for a two-group comparison divided by 3 (Bonferroni correction). In this case, the boundaries will be $Z=3.394$ for the interim analysis and $Z=2.400$ for the final analysis. Assuming that there are 30 subjects per group and that the standard deviation is 6.5 dB at the interim analysis, the boundary will be crossed if a group difference exceeds approximately 5.7 dB. This monitoring procedure will have a negligible impact on the overall Type I error probability: the significance level at the final analysis corresponding to $Z=2.400$ is $\alpha=0.0164$ . Point and interval estimates of treatment effects, as well as reported p-values, will be adjusted for the interim analysis. The bias-adjusted mean will be used for point estimation and confidence intervals and p-values based on the MLE (sample mean) ordering of the sample space defined by the group sequential design $^{97,98}$ will be reported in this case. |
| 1590<br>1591<br>1592<br>1593<br>1594<br>1595 | The efficacy boundary will be considered to be non-binding. We believe that it may be prudent to halt or modify the trial only if (1) two of the treatment groups are each shown to be superior to the third (in which case the third group may be dropped) or (2) one of the treatment groups is shown to be superior to each of the other two (in which case the trial may be halted). Of course, the relative safety profiles of the treatments would have to factor into these considerations as well. |
| 1596 | 9.9 Baseline Characteristics |
| 1597<br>1598<br>1599<br>1600 | Baseline characteristics of subjects will be summarized overall and by treatment group; formal statistical comparisons between treatment groups will not be performed. Continuous variables will be described using means, standard deviations, medians, quartiles, and ranges, and categorical variables will be described using percentages. |
| 1601 | 9.10 Sample Size Determination |
| 1602<br>1603<br>1604<br>1605<br>1606<br>1607 | In this clinical trial, 180 subjects with newly diagnosed IIH and moderate to severe visual loss ( $-27 \text{ dB} \le \text{PMD} \le -6 \text{ dB}$ ) will be randomly assigned to receive either medical therapy, ONSF + medical therapy, or VPS + medical therapy (60 per group). This sample size should provide high power to detect group differences when the true differences are of clinical significance, allowing for an anticipated 10% drop-out. The rationale for the choice of a clinically significant treatment group difference of 4.5 dB is explained in the last paragraph below. |
| 1608<br>1609<br>1610 | The primary outcome variable in this trial will be the change from baseline to the first of Month 6 or time of treatment failure in PMD in an eligible eye. An eye is defined as eligible if it satisfied the requirement of $-27 \text{ dB} \le \text{PMD} \le -6 \text{ dB}$ at baseline. The sample size considerations |

initially focus on data from the best eligible eye, since most subjects are expected to contribute only one eye to the primary analysis, but addition of the other eligible eye is also considered 1612 below. In 2012, the IIH Study Group performed a retrospective chart review of consecutive 1613 newly diagnosed patients that met the modified Dandy criteria for IIH<sup>27</sup> at 30 of the 41 1614 participating sites. Data on PMD were available from 91 patients at two time points, before and 1615 after intervention, with the median follow-up time being 6.0 months (interquartile range 4.1 to 1616 7.0 months). Patients received either medical treatment (n = 43), ONSF (n = 24), or VPS (n = 24), or 1618 24). The mean (± standard deviation) changes in PMD (in dB) in the best eligible eye over the follow-up period were  $5.5 \pm 6.9$  in the medical group,  $2.0 \pm 8.9$  in the ONSF group, and  $8.2 \pm 8.0$ 1619 1620 in the VPS group; overall these values were  $5.3 \pm 8.0$ . The distribution of these changes was slightly more peaked than would be expected for a normal distribution, as illustrated in Figure 4a 1622 and 4b.



Figure 4a and 4b. Distribution of Changes in PMD in the Best Eligible Eye

The figure on the left (a) shows the distribution of changes in PMD in the best eligible eye according to baseline PMD and intervention. Most of the patients demonstrated improvement in PMD. The figure on the right (b) shows a histogram of the changes in PMD in the best eligible eye regardless of intervention. The distribution appears to be characterized by a high concentration of changes between 0 and 10 PMD and is more peaked than normal.

Given the cross-sectional nature of the preliminary data, sample size determination based on the use of GEE for the primary analysis is very similar to that based on the use of an analysis of covariance model. If an analysis of covariance model is fit to the preliminary data, with change in PMD as the outcome variable and treatment group and baseline PMD as the independent variables, the standard deviation of the residuals is 6.3 dB. The differences between treatment groups in adjusted mean response are quite small in this analysis: -0.09 dB difference between the ONSF and medical groups, and 1.13 dB difference between the VPS and medical groups. Also, a GEE analysis produces identical adjusted group means and slightly different estimated standard errors than those from the analysis of covariance model.

1639 It may be noted that the standard deviation of the residuals in the above analysis of covariance 1640 model is substantially less than the standard deviations in the individual treatment groups. reflecting adjustment for the baseline value of PMD in the analysis of covariance model and the fairly strong correlation between the baseline and final PMD values (r = 0.52). When considering 1642

1611

1617

1621

1623

1624

1625

1626

1627

1628

1629

1630

1631

1632

1633

1634 1635

1636

1637 1638

1641

| 1643 | only subjects who were followed for at least $5.5$ months ( $n = 56$ ), the correlation between the |
|---|---|
| 1644 | baseline and final PMD values was actually somewhat higher ( $r = 0.62$ ) and the residual standard |
| 1645 | deviation in the analysis of covariance model was smaller (6.0 dB). |
| 1646 | Assuming a standard deviation of 6.5 dB, consistent with the preliminary data, and a Bonferroni- |
| 1647 | adjusted two-tailed significance level of 1.7%, in order to detect a group difference assuming a |
| 1648 | true difference of 4.5 dB with 88% power, a sample size of 54 subjects per group is required. |
| 1649 | The sample size will be inflated to 60 subjects per group (180 total) to accommodate an |
| 1650 | anticipated 10% rate of subject withdrawal/dropout. The power remains above 80% even if the |
| 1651 | assumed standard deviation is as large as 7.1 dB. |
| 1652 | The inclusion of the worst eligible eye is expected to increase power, but the increase is expected |
| 1653 | to be small (approximately 3%) because the preliminary data from the chart review indicate that |
| 1654 | only ~40% of subjects will contribute a second eligible eye to the analysis and the correlation |
| 1655 | between the outcomes in the two eyes is quite high (0.82 in our sample). This assumes that the |
| 1656 | group difference will be comparable in the best and worst eligible eyes, as we anticipate. |
| 1657 | The chosen effect size of 4.5 dB is based on the following rationale. Visual field defects are |
| 1658 | similar in IIH and glaucoma <sup>1,85</sup> and data on the relationship between vision-specific quality of |
| 1659 | life (as measured by the NEI-VFQ-25) and PMD from the better seeing eye are available from |
| 1660 | 213 subjects with glaucoma in the Los Angeles Latino Eye Study <sup>86</sup> . A regression analysis |
| 1661 | yielded the finding that a change of 1 dB in PMD corresponded to an approximately one-unit |
| 1662 | score change on the NEI-VFQ-25 composite score. 86,87 In another study, Suner et al. used data |
| 1663 | from two clinical trials in neovascular age-related macular degeneration and anchor-based |
| 1664 | methods to estimate the change in NEI-VFQ-25 composite score that corresponds to a change of |
| 1665 | ≥ 15 letters (~ 3 lines) in visual acuity, a value generally accepted as clinically significant. <sup>87</sup> |
| 1666 | They concluded that a change of 4-6 points on the NEI-VFQ-25 composite score should be |
| 1667 | considered clinically significant. Taken together, the results of these two investigations suggest |
| 1668 | that a change in PMD of 4.5 dB corresponds to a change in NEI-VFQ-25 score that would be |
| 1669 | considered to be of minimal clinical significance. |
| 1670 | |
| 1671 | <b>Chapter 10: Data Collection and Monitoring</b> |
|---|---|
| 1672 | 10.1 Case Report Forms |
| 1673<br>1674 | The main study data are collected through electronic case report forms (CRFs). These electronic CRFs from the study website are considered the primary source documentation. |
| 1675<br>1676<br>1677<br>1678 | When data are directly collected in electronic case report forms, this will be considered the source data. Each participating site will maintain appropriate medical and research records for this trial, in compliance with ICH E6 and regulatory and institutional requirements for the protection of confidentiality of subjects. |
| 1679 | 10.2 Study Records Retention |
| 1680<br>1681<br>1682<br>1683<br>1684 | Study documents should be retained for a minimum of 3 years in accordance with NIH and FDA requirements. These documents should be retained for a longer period, however, if required by local regulations. No records will be destroyed without the written consent of the sponsor, if applicable. It is the responsibility of the sponsor to inform the investigator when these documents no longer need to be retained. |
| 1685 | 10.3 Quality Assurance and Monitoring |
| 1686<br>1687<br>1688<br>1689<br>1690 | Designated personnel from the Coordinating Center will be responsible for maintaining quality assurance (QA) and quality control (QC) systems to ensure that the clinical portion of the trial is conducted and data are generated, documented and reported in compliance with the protocol, Good Clinical Practice (GCP) and the applicable regulatory requirements. Adverse events will be prioritized for monitoring. |
| 1691<br>1692<br>1693<br>1694 | A risk-based monitoring (RBM) plan will be developed and revised as needed during the course of the study, consistent with the FDA "Guidance for Industry Oversight of Clinical Investigations — A Risk-Based Approach to Monitoring" (August 2013). Study conduct and monitoring will conform with 21 Code of Federal Regulations (CFR) 312. |
| 1695<br>1696<br>1697<br>1698 | The data of most importance for monitoring at the site are subject eligibility and adverse events. Therefore, the RBM plan will focus on these areas. As much as possible, remote monitoring will be performed in real-time with on-site monitoring performed to evaluate the verity and completeness of the key site data. Elements of the RBM may include: |
| 1699 | • Qualification assessment, training, and certification for sites and site personnel |
| 1700<br>1701 | <ul> <li>Oversight of Institutional Review Board (IRB) coverage and informed consent procedures</li> </ul> |
| 1702<br>1703 | • Central (remote) data monitoring: validation of data entry, data edits/audit trail, protocol review of entered data and edits, statistical monitoring, study closeout |
| 1704 | • On-site monitoring (site visits): source data verification, site visit report |
| 1705 | Agent/Device accountability |
| 1706 | Communications with site staff |

| 1707 | Patient retention and visit completion |
|---|---|
| 1708 | Quality control reports |
| 1709 | Management of noncompliance |
| 1710 | <ul> <li>Documenting monitoring activities</li> </ul> |
| 1711 | Adverse event reporting and monitoring |
| 1712<br>1713<br>1714<br>1715 | Coordinating Center representatives or their designees may visit the study facilities at any time in order to maintain current and personal knowledge of the study through review of the records, comparison with source documents, observation and discussion of the conduct and progress of the study. |
| 1716 | 10.4 Protocol Deviations |
| 1717<br>1718<br>1719<br>1720 | A protocol deviation is any noncompliance with the clinical trial protocol, GCP, or procedure requirements. The noncompliance may be either on the part of the subject, the investigator, or the study site staff. As a result of deviations, corrective actions are to be developed by the site and implemented promptly. |
| 1721<br>1722 | The site PI/study staff is responsible for knowing and adhering to their IRB requirements. Further details about the handling of protocol deviations will be included in the monitoring plan. |
| 1723 | 10.5 Committees and Reading Centers |
| 1724 | 10.5.1 Resource Center (RC) |
| 1725<br>1726<br>1727<br>1728 | The Resource Center at Mount Sinai will oversee all three reading centers described below. The Resource Center will review quarterly quality control reports. Calls and on-site monitoring visits will be conducted as necessary to address substandard performance. The RC will also assist the reading centers in analyses of visual fields, fundus photos, and OCT images as needed. |
| 1729 | 10.5.2 Visual Field Reading Center (VFRC) |
| 1730<br>1731<br>1732<br>1733<br>1734 | The Iowa VFRC will provide training and certification of all technicians (at least 2 per clinic site) so that valid perimetry results are transmitted, read, stored and archived. They will also provide ongoing analysis of the primary outcome variable, perimetric mean deviation (PMD) to the sites, Jaeb Center, RC, Adjudication Committee, Surgical Malfunction Review Committee and SSC. |
| 1735<br>1736<br>1737<br>1738 | Sites will upload Humphrey Field Analyzer size V Full Threshold native data files using the secure VFRC upload facility. The VFRC will then generate a size V "Statpac"-like pdf printout with the necessary statistical indices and transfer the pdf back to the site for all valid submitted visual field examinations. |
| 1739<br>1740 | Data will be stored on a secure server. Daily, weekly and monthly backups of the data will be made with offsite storage as well. |

| 1741<br>1742 | Each examination will have quality control checks for internal validity. Monthly and quarterly quality control reports will be generated for the RC and SSC. |
|---|---|
| 1743 | 10.5.3 Photographic Reading Center (PRC) |
| 1744<br>1745<br>1746<br>1747 | The Rochester PRC will provide training and certification of all technicians (at least 1 per clinic site) so that valid photographic images are transmitted, read, stored and archived. They will also provide ongoing grading of the photos to the sites, Jaeb Center, RC, Adjudication Committee, Surgical Malfunction Review Committee and SSC. |
| 1748<br>1749<br>1750 | Fundus photos will be transferred to the PRC from the site via a secure file transfer upload client. Each site will be given an internal address and password that allows the site to upload subject images. |
| 1751<br>1752 | Data will be stored on a secure server. Daily, weekly and monthly backups of the data will be made with offsite storage as well. Quality Control reports will be prepared on a quarterly basis. |
| 1753 | 10.5.4 Optical Coherence Tomography Reading Center (OCTRC) |
| 1754<br>1755<br>1756<br>1757<br>1758 | The OCTRC will provide training and certification of all technicians (at least 1 per clinic site) so that valid OCT images are transmitted, read, stored and archived. They will also provide ongoing assessment of thickness measurements and evaluation of the optic nerve head neural canal shape deformations to the sites, Jaeb Center, RC, Adjudication Committee, Surgical Malfunction Review Committee and SSC. |
| 1759<br>1760<br>1761 | Raw data will be transferred to the OCTRC from the site via UC Davis OCTRC's secure File Transfer Protocol (FTP) site. These raw data will be uploaded into the Cirrus Research Browser for assessment and quality control by the OCTRC. |
| 1762<br>1763<br>1764 | Data will be stored on a secure server. Daily, weekly and monthly backups of the data will be made with offsite storage as well. Quality control reports will be produced by the OCTRC on a quarterly basis. |
| 1765 | 10.5.5 Surgical Quality Assurance Committee (SQAC) |
| 1766<br>1767 | There will be a SQAC composed of two orbital surgeons and two neurosurgeons. They will certify study surgeons and provide quality control, as detailed in the MOP. |
| 1768 | 10.5.6 Surgical Malfunction Review Committee (SMRC) |
| 1769<br>1770<br>1771 | The SMRC will review patients in the trial that are worsening and determine if possible surgical malfunction exists. The review is triggered if the criteria described in section 5.6.1 above are met. |

| 1772 | 10.5.7 Adjudication Committee (AC) |
|---|---|
| 773 | A three member committee appointed by the Study Steering Committee (SSC), plus the Study |
| 774 | Director, will review subjects that meet the criteria for possible treatment failure. All treatment |
| 775 | failure cases will be reviewed first by the Study Director or committee chair for safety reasons. |
| 776 | This committee will be charged with deciding whether the worsening of the subject is most |
| 777 | likely due to increased intracranial pressure and is a failure of therapy, or the worsening of PMD |
| 778 | is more likely due to another reason. A report of all decisions will be sent to the Data and Safety |
| 779 | Monitoring Committee (DSMC). Records of visual fields, fundus photos, and OCTs will be |
| 780 | provided to the coordinating center to organize with the clinical information for use by the Study |
| 781 | Director and AC. |

| 1782 | Chapter 11: Ethics/Protection of Human Subjects |
|---|---|
| 1783 | 11.1 Ethical Standard |
| 1784 | The investigator will ensure that this study is conducted in full conformity with Regulations for |
| 1785 | the Protection of Human Subjects of Research codified in 45 CFR Part 46, 21 CFR Part 50, 21 |
| 1786 | CFR Part 56, and/or the ICH E6. |
| 1787 | 11.2 Institutional Review Boards |
| 1788 | The protocol, informed consent form(s), recruitment materials, and all participant materials will |
| 1789 | be submitted to the IRB for review and approval. Approval of both the protocol and the consent |
| 1790 | form must be obtained before any subject is enrolled. Any amendment to the protocol will |
| 1791 | require review and approval by the IRB before the changes are implemented to the study. All |
| 1792 | changes to the consent form will be IRB approved; a determination will be made regarding |
| 1793 | whether previously consented subjects need to be re-consented. |
| 1794 | 11.3 Informed Consent Process |
| 1795 | 11.3.1 Consent Procedures and Documentation |
| 1796 | Informed consent is a process that is initiated prior to the individual's agreeing to participate in |
| 1797 | the study and continues throughout the individual's study participation. Extensive discussion of |
| 1798 | risks and possible benefits of participation will be provided to the subjects and their families. |
| 1799 | Consent forms will be IRB-approved and the subject will be asked to read and review the |
| 1800 | document. The investigator will explain the research study to the subject and answer any |
| 1801 | questions that may arise. All subjects will receive a verbal explanation in terms suited to their |
| 1802 | comprehension of the purposes, procedures, and potential risks of the study and of their rights as |
| 1803 | research subjects. Subjects will have the opportunity to carefully review the written consent |
| 1804 | form and ask questions prior to signing. |
| 1805 | The subjects should have the opportunity to discuss the study with their surrogates or think about |
| 1806 | it prior to agreeing to participate. The subject will sign the informed consent document prior to |
| 1807 | any procedures being done specifically for the study. The subjects may withdraw consent at any |
| 1808 | time throughout the course of the trial. A copy of the informed consent document will be given |
| 1809 | to the subjects for their records. The rights and welfare of the subjects will be protected by |
| 1810 | emphasizing to them that the quality of their medical care will not be adversely affected if they |
| 1811 | decline to participate in this study. |
| 1812 | 11.3.2 Subject and Data Confidentiality |
| 1813 | Subject confidentiality is strictly held in trust by the participating investigators, their staff, the |
| 1814 | coordinating center, reading centers, and their agents. This confidentiality is extended to cover |
| 1815 | testing of biological samples and genetic tests in addition to the clinical information relating to |
| 1816 | subjects. Therefore, the study protocol, documentation, data, and all other information generated |
| 1817 | will be held in strict confidence. No information concerning the study or the data will be |
| 1818 | released to any unauthorized third party without prior written approval of NORDIC. |

| 1819<br>1820<br>1821<br>1822<br>1823 | The study monitor, other authorized representatives of the coordinating center and NORDIC, and representatives of the IRB may inspect all documents and records required to be maintained by the investigator, including but not limited to, medical records (office, clinic, or hospital) and pharmacy records for the subjects in this study. The clinical study site will permit access to such records. |
|---|---|
| 1824<br>1825<br>1826<br>1827 | The study subject's contact information will be securely stored at each clinical site for internal use during the study. At the end of the study, all records will continue to be kept in a secure location for as long a period as dictated by IRB, NIH, other regulatory bodies, and institutional regulations. |
| 1828<br>1829<br>1830<br>1831<br>1832<br>1833<br>1834<br>1835<br>1836<br>1837 | Visual field data will be transmitted to the VFRC at the University of Iowa, OCT image data will be transmitted to the University of California at Davis Reading Center, and optic disc photographs will be transmitted to the Photographic Reading Center at the University of Rochester. These data will not include the subject's contact or identifying information. Rather, individual subjects and their research data will be identified by a unique study identification number. All study subject research data, which is for purposes of statistical analysis and scientific reporting, will be transmitted to and stored at the Jaeb Center for Health Research. The study data entry and study management systems used by clinical sites and by the Jaeb Center research staff will be secured and password protected. At the end of the study, all study databases will be de-identified and placed in the public domain by the Jaeb Center. |
| 1838<br>1839<br>1840<br>1841<br>1842<br>1843<br>1844<br>1845 | The Certificate of Confidentiality provided by NIH further protects the privacy of study subjects. This certificate protects identifiable research information from forced disclosure. It allows the investigator and others who have access to research records to refuse to disclose identifying information on research participation in any civil, criminal, administrative, legislative, or other proceeding, whether at the federal, state, or local level. By protecting researchers and institutions from being compelled to disclose information that would identify research subjects, Certificates of Confidentiality help achieve the research objectives and promote participation in studies by helping assure confidentiality and privacy to subjects. |
| 1846 | 11.3.3 Future Use of Stored Specimens |
| 1847<br>1848<br>1849 | Permission to collect and store blood samples for future use will be included in the informed consent. With the subject's approval, blood specimens will be labeled by study ID and stored in a central lab for use by researchers, including those outside of the study. |
| 1850<br>1851<br>1852 | These samples could be used for research such as metabolomics studies on lipid and proteins, which include gender and obesity hormones, and microRNA for specific proteins or autoimmune factors. |
| 1853<br>1854<br>1855 | All studies will be performed after a written protocol for testing and analysis are approved by the study steering committee and local IRB(s). Specimens will be transferred to research labs at research institutions as needed to perform the approved investigations. |
| 1856<br>1857<br>1858 | The central lab will also be provided with a code-link for each subject that will allow linking the biological specimens with the clinical information collected during the trial, maintaining the masking of the identity of the subject. |

| 1859 | During the conduct of the study, an individual subject can choose to withdraw consent to have |
|---|---|
| 1860 | biological specimens stored for future research. However, withdrawal of consent with regard to |
| 1861 | biosample storage will not be possible after the study is completed. |

# 1862 Chapter 12: References

- 1863 1. Wall, M and George, D. Idiopathic intracranial hypertension. A prospective study of 50 patients. Brain. 1991; 114:155-180.
- Wall, M, McDermott, MP, Kieburtz, KD, et al. Effect of acetazolamide on visual function in patients with idiopathic intracranial hypertension and mild visual loss: the idiopathic intracranial hypertension treatment trial. JAMA. 2014;1641-1651.
- Hayreh, SS. Pathogenesis of oedema of the optic disc (papilloedema): a preliminary report. Br J Ophthalmol. 1964; 48:522-542.
- 1870 4. Smith, JL, Hoyt, WF, and Newton, TH. Optic nerve sheath decompression for relief of chronic monocular choked disc. Am J Ophthalmol. 1969; 68:633-639.
- 1872 5. Corbett, JJ, Nerad, JA, Tse, DT, et al. Results of optic nerve sheath fenestration for pseudotumor cerebri. The lateral orbitotomy approach. Arch Ophthalmol. 1988; 106:1391-1397.
- Hamed, LM, Tse, DT, Glaser, JS, et al. Neuroimaging of the optic nerve after fenestration for management of pseudotumor cerebri. Arch Ophthalmol. 1992; 110:636-639.
- 7. Yazici, Z, Yazici, B, and Tuncel, E. Findings of magnetic resonance imaging after optic nerve sheath decompression in patients with idiopathic intracranial hypertension. Am J Ophthalmol. 2007; 144:429-435.
- 1880 8. Keltner, JL, Albert, DA, Lubow, M, et al. Optic nerve decompression. A clinical pathologic study. Arch Ophthalmol. 1977; 95:97-104.
- 9. Smith, CH and Orcutt, JC. Surgical treatment of pseudotumor cerebri. Int Ophthalmol Clin. 1883 1986; 26:265-275.
- 1884 10. Killer, HE, Jaggi, GP, Flammer, J, et al. Cerebrospinal fluid dynamics between the intracranial and the subarachnoid space of the optic nerve. Is it always bidirectional? Brain. 2007; 130:514-520.
- 1887 11. Wilkes, BN and Siatkowski, RM. Progressive optic neuropathy in idiopathic intracranial hypertension after optic nerve sheath fenestration. J Neuroophthalmol. 2009;281-283.
- 1889 12. Spoor, TC and McHenry, JG. Long-term effectiveness of optic nerve sheath decompression for pseudotumor cerebri. Arch Ophthalmol. 1993; 111:632-635.
- 1891 13. Wall, M, Johnson, CA, Kutzko, KS, et al. Long- and short-term variability of automated perimetry results in patients with optic neuritis and healthy subjects. Arch Ophthalmol. 1998;53-61.
- 1894 14. Johnston, I, Besser, M, and Morgan, MK. Cerebrospinal fluid diversion in the treatment of benign intracranial hypertension. J Neurosurg. 1988; 69:195-202.

- 1896 15. Burgett, RA, Purvin, VA, and Kawasaki, A. Lumboperitoneal shunting for pseudotumor cerebri. Neurology. 1997; 49:734-739.
- 1898 16. Eggenberger, ER, Miller, NR, and Vitale, S. Lumboperitoneal shunt for the treatment of pseudotumor cerebri. Neurology. 1996; 46:1524-1530.
- 1900 17. Rosenberg, M, Smith, C, and Beck, R. The efficacy of shunting procedures in pseudotumor cerebri. Neurology. 1989; 39:209.
- 1902 18. Karabatsou, K, Quigley, G, Buxton, N, et al. Lumboperitoneal shunts: are the complications acceptable? Acta Neurochirurgica 146(11):1193-7. 2004.
- 19. McGirt, MJ, Woodworth, G, Thomas, G, et al. Cerebrospinal fluid shunt placement for pseudotumor cerebri-associated intractable headache: predictors of treatment response and an analysis of long-term outcomes. Journal of Neurosurgery 101(4):627-32. 2004.
- 1907 20. Bynke, G, Zemack, G, Bynke, H, et al. Ventriculoperitoneal shunting for idiopathic intracranial hypertension. Neurology 63(7):1314-6. 2004.
- 1909 21. Abubaker, K, Ali, Z, Raza, K, et al. Idiopathic intracranial hypertension: lumboperitoneal shunts versus ventriculoperitoneal shunts--case series and literature review. Br J Neurosurg. 2011; 25:94-99.
- 1912 22. Tarnaris, A, Toma, AK, Watkins, LD, et al. Is there a difference in outcomes of patients with idiopathic intracranial hypertension with the choice of cerebrospinal fluid diversion site: a single centre experience. Clin Neurol Neurosurg. 2011; 113:477-479.
- Lueck, C and McIllwaine, G. Interventions for Idiopathic Intracranial Hypertension. The
   Cochrane Library. 2009;1-10.
- 1917 24. Piper, RJ, Kalyvas, AV, Young, AM, et al. Interventions for idiopathic intracranial hypertension. Cochrane Database Syst Rev. 2015;CD003434.
- 1919 25. Curry, WT, Jr., Butler, WE, and Barker, FG. Rapidly rising incidence of cerebrospinal fluid 1920 shunting procedures for idiopathic intracranial hypertension in the United States, 1988-1921 2002. Neurosurgery 57(1):97-108; discussion 97-108. 2005.
- 1922 26. Friesner, D, Rosenman, R, Lobb, BM, et al. Idiopathic intracranial hypertension in the USA: the role of obesity in establishing prevalence and healthcare costs. Obes Rev. 2011; 12:e372-e380.
- 1925 27. Smith, JL. Whence pseudotumor cerebri? J Clin Neuro-ophthalmol. 1985; 5:55-56.
- Wall, M, Kutzko, KS, and Chauhan, BC. Variability in patients with glaucomatous optic
   nerve damage is reduced using size V stimuli. Invest Ophthalmol Vis Sci. 1997; 38:426 435.

- 1929 29. Wall, M, Woodward, KR, Doyle, CK, et al. Repeatability of automated perimetry: a comparison between standard automated perimetry with stimulus size III and V, matrix, and motion perimetry. Invest Ophthalmol Vis Sci. 2009; 50:974-979.
- 1932 30. Wall, M, Woodward, KR, Doyle, CK, et al. The effective dynamic ranges of standard automated perimetry sizes III and V and motion and matrix perimetry. Arch Ophthalmol. 2010; 128:570-576.
- 1935 31. Berson, EL, Rosner, B, Sandberg, MA, et al. Clinical trial of lutein in patients with retinitis pigmentosa receiving vitamin A. Arch Ophthalmol. 2010; 128:403-411.
- 32. Gardiner, SK, Swanson, WH, Goren, D, et al. Assessment of the Reliability of Standard
   Automated Perimetry in Regions of Glaucomatous Damage. Ophthalmology. 2014;10.
- 1939 33. Swanson, WH, Felius, J, and Birch, DG. Effect of stimulus size on static visual fields in patients with retinitis pigmentosa. Ophthalmology. 2000; 107:1950-1954.
- 34. Swanson, WH. Stimulus size for perimetry in patients with glaucoma. Invest Ophthalmol
   Vis Sci. 2013; 54:3984-12335.
- 35. Swanson, WH, Dul, MW, Horner, DG, et al. Assessing spatial and temporal properties of
   perimetric stimuli for resistance to clinical variations in retinal illumination. Invest
   Ophthalmol Vis Sci. 2014; %20;55:353-359.
- 1946 36. Wall, M, Doyle, CK, Zamba, KD, et al. The repeatability of mean defect with size III and size V standard automated perimetry. Invest Ophthalmol Vis Sci. 2013; 54:1345-1351.
- 1948 37. Papilledema Outcomes from the Optical Coherence Tomography Substudy of the Idiopathic Intracranial Hypertension Treatment Trial. Ophthalmology. 2015; 122:1939-1945.
- 38. Wang JK, Kardon R, Ledholter J, Sibony P, Kupersmith M, Garvin M, on behalf of the
   OCT Sub-Study Committee for the NORDIC Idiopathic Intracranial Hypertension Study
   Group. Peripapillary Retinal Pigment Epithelium Layer Shape Changes from Acetazolamide
   Treatment in the Idiopathic Intracranial Hypertension Treatment Trial. IOVS 2017;58:2554-
- 1954 265. doi:10.1167/iovs.16-21089
- 39. Sibony, P, Kupersmith, MJ, and Rohlf, FJ. Shape analysis of the peripapillary RPE layer in papilledema and ischemic optic neuropathy. Invest Ophthalmol Vis Sci. 2011; 52:7987-7995.
- 1958 40. Chen, JJ, Thurtell, MJ, Longmuir, RA, et al. Causes and Prognosis of Visual Acuity Loss at
   1959 the Time of Initial Presentation in Idiopathic Intracranial Hypertension. Invest Ophthalmol
   1960 Vis Sci. 2015; 56:3850-3859.
- 1961 41. Skelton J, Beech B. Attrition in paediatric weight management: a review of the literature and new directions. Obesity Reviews 2011;12, e273-e281

- 1963 42. Schoeman, J, Donald, P, van Zyl, L, et al. Tuberculous hydrocephalus: comparison of different treatments with regard to ICP, ventricular size and clinical outcome.
- Developmental Medicine & Child Neurology. 1991; 33:396-405.
- 43. Schoeman, JF. Childhood pseudotumor cerebri: clinical and intracranial pressure response
   to acetazolamide and furosemide treatment in a case series. J Child Neurol. 1994; 9:130 134.
- 44. Schoeman, JF, Honey, EM, and Loock, DB. Raised ICP in a child with cryptococcal
   meningitis: CT evidence of a distal CSF block. Childs Nervous System. 1996; 12:568-571.
- 1971 45. Kupersmith, MJ, Gamell, L, Turbin, R, et al. Effects of weight loss on the course of idiopathic intracranial hypertension in women. Neurology. 1998; 50:1094-1098.
- 1973 46. Johnson, LN, Krohel, GB, Madsen, RW, et al. The role of weight loss and acetazolamide in 1974 the treatment of idiopathic intracranial hypertension (pseudotumor cerebri). Ophthalmology. 1975 1998; 105:2313-2317.
- 1976 47. Hupp, SL, Glaser, JS, and Frazier-Byrne, S. Optic nerve sheath decompression. Review of 1977 17 cases. Arch Ophthalmol. 1987; 105:386-389.
- 48. Sergott, RC, Savino, PJ, and Bosley, TM. Modified optic nerve sheath decompression
   provides long-term visual improvement for pseudotumor cerebri. Arch Ophthalmol. 1988;
   106:1391-1397.
- 49. Brourman, ND, Spoor, TC, and Ramocki, JM. Optic nerve sheath decompression for pseudotumor cerebri. Arch Ophthalmol. 1988; 106:1378-1383.
- 1983 50. Goh, KY, Schatz, NJ, and Glaser, JS. Optic nerve sheath fenestration for pseudotumor cerebri. J Neuro-Ophthalmol. 1997; 17:86-91.
- 1985 51. Plotnik, JL and Kosmorsky, GS. Operative complications of optic nerve sheath decompression. Ophthalmology. 1993; 100:683-690.
- 1987 52. Acheson, JF, Green, WT, and Sanders, MD. Optic nerve sheath decompression for the 1988 treatment of visual failure in chronic raised intracranial pressure. J Neurol Neurosurg 1989 Psychiatr. 1994; 57:1426-1429.
- 1990 53. Kelman, SE, Heaps, R, Wolf, A, et al. Optic nerve decompression surgery improves visual function in patients with pseudotumor cerebri. Neurosurgery. 1992; 30:391-395.
- 1992 54. Banta, JT and Farris, BK. Pseudotumor cerebri and optic nerve sheath decompression.
   1993 Ophthalmology. 2000; 107:1907-1912.
- 1994 55. Alsuhaibani, AH, Carter, KD, Nerad, JA, et al. Effect of optic nerve sheath fenestration on papilledema of the operated and the contralateral nonoperated eyes in idiopathic intracranial hypertension. Ophthalmology. 2011; 118:412-414.

- 1997 56. Pineles, S and Volpe, N. Long-Term Results of Optic Nerve Sheath Fenestration for Idiopathic Intracranial Hypertension: Earlier Intervention Favours Improved Outcomes.
- 1999 Neuro-Ophthalmology. 2013; 37:12-19.
- 57. Fonseca, PL, Rigamonti, D, Miller, NR, et al. Visual outcomes of surgical intervention for pseudotumour cerebri: optic nerve sheath fenestration versus cerebrospinal fluid diversion.
   Br J Ophthalmol. 2014; 98:1360-1363.
- 2003 58. Rosenberg, ML, Corbett, JJ, Smith, C, et al. Cerebrospinal fluid diversion procedures in pseudotumor cerebri. Neurology. 1993; 43:1071-1072.
- 59. Shapiro, S, Yee, R, and Brown, H. Surgical management of pseudotumor cerebri in pregnancy: case report. Neurosurgery. 1995; 37:829-831.
- Tulipan, N, Lavin, PJ, and Copeland, M. Stereotactic ventriculoperitoneal shunt for
   idiopathic intracranial hypertension: technical note. Neurosurgery. 2009; discussion 176-7.: 7.
- 2010 61. Maher, CO, Garrity, JA, and Meyer, FB. Refractory idiopathic intracranial hypertension treated with stereotactically planned ventriculoperitoneal shunt placement. Neurosurg Focus. 2001; 10:E1.
- 2013 62. Abu-Serieh, B, Ghassempour, K, Duprez, T, et al. Stereotactic ventriculoperitoneal shunting for refractory idiopathic intracranial hypertension. Neurosurgery. 2007; 60:1039-1043.
- 2016 63. Nadkarni, TD, Rekate, HL, and Wallace, D. Concurrent use of a lumboperitoneal shunt with programmable valve and ventricular access device in the treatment of pseudotumor cerebri: review of 40 cases. J Neurosurg Pediatr. 2008; 2:19-24.
- Kandasamy, J, Hayhurst, C, Clark, S, et al. Electromagnetic stereotactic
   ventriculoperitoneal CSF shunting for idiopathic intracranial hypertension: a successful step
   forward? World Neurosurg. 2011 Jan; 75(1):155-60; discussion 32-3.
- 2022 65. Sinclair, AJ, Kuruvath, S, Sen, D, et al. Is cerebrospinal fluid shunting in idiopathic intracranial hypertension worthwhile? A 10-year review. Cephalalgia. 2011; 31:1627-1633.
- 2024 66. El-Saadany, WF, Farhoud, A, and Zidan, I. Lumboperitoneal shunt for idiopathic intracranial hypertension: patients' selection and outcome. Neurosurg Rev. 2012; 35:239-243.
- 2027 67. Yadav, YR, Parihar, V, Agarwal, M, et al. Lumbar peritoneal shunt in idiopathic intracranial hypertension. Turk Neurosurg. 2012; 22:21-26.
- Huang, LC, Winter, TW, Herro, AM, et al. Ventriculoperitoneal shunt as a treatment of visual loss in idiopathic intracranial hypertension. J Neuroophthalmol. 2014; 34:223-228.

- 2031 69. Rizzo, JL, Lam, KV, Wall, M, et al. Perimetry, Retinal Nerve Fiber Layer Thickness and
- 2032 Papilledema Grade After Cerebrospinal Fluid Shunting in Patients With Idiopathic
- 2033 Intracranial Hypertension. J Neuroophthalmol. 2014.
- 70. Farb, RI, Vanek, I, Scott, JN, et al. Idiopathic intracranial hypertension: the prevalence and
- morphology of sinovenous stenosis. Neurology. 2003; 60:1418-1424.
- 2036 71. Wall, M, Kupersmith, MJ, Kieburtz, KD, et al. The Idiopathic Intracranial Hypertension
- Treatment Trial: Clinical Profile at Baseline. JAMA Neurol doi: 10 1001/jamaneurol 133.
- 2038 2014.
- 2039 72. Lee, AG, Anderson, R, Kardon, RH, et al. Presumed "sulfa allergy" in patients with
- intracranial hypertension treated with acetazolamide or furosemide: cross-reactivity, myth or
- 2041 reality? Am J Ophthalmol. 2004; 138:114-118.
- 2042 73. Epstein, DL and Grant, WM. Carbonic anhydrase inhibitor side effects. Serum chemical
- analysis. Arch Ophthalmol. 1977; 95:1378-1382.
- 2044 74. Zimran, A and Beutler, E. Can the risk of acetazolamide-induced aplastic anemia be
- decreased by periodic monitoring of blood cell counts? Am J Ophthalmol. 1987; 104:654-
- 2046 658.
- 2047 75. Mogk, LG and Cyrlin, MN. Blood dyscrasias and carbonic anhydrase inhibitors.
- 2048 Ophthalmology. 1988; 95:768-771.
- 2049 76. Wall, M and White, WN. Asymmetric papilledema in idiopathic intracranial hypertension:
- prospective interocular comparison of sensory visual function. Invest Ophthalmol Vis Sci.
- 2051 1998; 39:134-142.
- 2052 77. Frisén, L. Swelling of the optic nerve head: a staging scheme. J Neurol Neurosurg Psychiatr.
- 2053 1982; 45:13-18.
- 2054 78. Scott, CJ, Kardon, RH, Lee, AG, et al. Diagnosis and grading of papilledema in patients
- with raised intracranial pressure using optical coherence tomography vs clinical expert
- assessment using a clinical staging scale. Arch Ophthalmol. 2010;705-711.
- 2057 79. Kleinschmidt, JJ, Digre, KB, and Hanover, R. Idiopathic intracranial hypertension:
- relationship to depression, anxiety, and quality of life. Neurology. 2000; 54:319-324.
- 2059 80. Kosinski, M, Bayliss, MS, Bjorner, JB, et al. A six-item short-form survey for measuring
- 2060 headache impact: the HIT-6. Qual Life Res. 2003; 12:963-974.
- 2061 81. Orcutt, JC, Page, NG, and Sanders, MD. Factors affecting visual loss in benign intracranial
- 2062 hypertension. Ophthalmology. 1984; 91:1303-1312.
- 2063 82. Wall, M. The headache profile of idiopathic intracranial hypertension. Cephalalgia. 1990;
- 2064 10:331-335.

- 2065 83. Friedman, DI and Rausch, EA. Headache diagnoses in patients with treated idiopathic intracranial hypertension. Neurology. 2002; 58:1551-1553.
- 2067 84. Efron, B and Tibshirani, RJ. An Introduction to Bootstrap. Chapter 25. Boca Raton, FL: Chapman and Hall / CRC, 1993.
- 2069 85. Grehn, F, Knorr-Held, S, and Kommerell, G. Glaucomatous like visual field defects in chronic papilledema. Albrecht von Graefes Arch Klin Exp Ophthalmol. 1981; 217:99-109.
- 2071 86. McKean-Cowdin, R, Wang, Y, Wu, J, et al. Impact of visual field loss on health-related quality of life in glaucoma: the Los Angeles Latino Eye Study. Ophthalmology. 2008; 115:941-948.
- 2074 87. Suner, IJ, Kokame, GT, Yu, E, et al. Responsiveness of NEI VFQ-25 to changes in visual acuity in neovascular AMD: validation studies from two phase 3 clinical trials. Invest Ophthalmol Vis Sci. 2009; 50:3629-3635.
- 88. Molenberghs, G and Kenward, MG. Missing Data in Clinical Studies. Chichester, UK: John Wiley and Sons, 2007.
- 2079 89. Little, RJA and Rubin, DB. Statistical Analysis with Missing Data. Second ed. Hoboken: John Wiley and Sons, 2002.
- 2081 90. D'Agostino, RB, Jr. Propensity score methods for bias reduction in the comparison of a treatment to a non-randomized control group. Stat Med. 1998; 17:2265-2281.
- 2083 91. Lunceford, JK and Davidian, M. Stratification and weighting via the propensity score in estimation of causal treatment effects: a comparative study. Stat Med. 2004; 23:2937-2960.
- 2085 92. Molenberghs, G, Thijs, H, Jansen, I, et al. Analyzing incomplete longitudinal clinical trial data. Biostatistics. 2004; 5:445-464.
- 208793. Rubin, DB. Multiple Imputation for Nonresponse in Surveys. New York: John Wiley and2088Sons, 1987.
- 2089 94. Reiter, JP and Raghunathan, TE. The multiple adaptations of multiple imputation. J Am Statist Asso. 2007; 102:1462-1471.
- 2091 95. Li KH. Imputation using Markov chains. Journal of Statistical Computation and Simulation. 1988; 30(1):57-79.
- 2093 96. Liu C. Bartlett's Decomposition of the Posterior Distribution of the Covariance for Normal Monotone Ignorable Missing Data. Journal of Multivariate Analysis. 1993;46(2):198–206.
- 2095 97. Cook TD, DeMets DL. Introduction to statistical methods for clinical trials. Boca Raton: Chapman & Hall/CRC; 2008.

- 98. Jennison C, Turnbull BW. Group sequential methods with applications to clinical trials.
   Boca Raton: Chapman & Hall/CRC; 2000.
- 2099 99. Follmann, DA, Proschan, MA, and Geller, NL. Monitoring pairwise comparisons in multi-2100 armed clinical trials. Biometrics. 1994; 50:325-336.
- 100. Cole SR, Hernán MA, Margolick JB, Cohen MH, Robins JM. Marginal structural models
   for estimating the effect of highly active antiretroviral therapy initiation on CD4 cell count.
   Am J Epidemiol 2005; 162:471-478.
- 2104 101. Grambsch PM, Therneau TM. Proportional hazards tests and diagnostics based on weighted residuals. Biometrika 1994; 81:515-526.
- 2106 102. Hosmer DW Jr., Lemeshow S. Applied Survival Analysis. New York NY: John Wiley and Sons, 1999.
- 2108 103. Kalbfleisch JD, Prentice RL. The Statistical Analysis of Failure Time Data, Second Edition.
   2109 Hoboken, NJ: John Wiley and Sons, 2002.
- 2110 104. Robins JM, Hernán MA, Brumback B. Marginal structural models and causal inference in epidemiology. Epidemiology 2000; 11:550-560.